CLINICAL TRIAL: NCT04895982
Title: A PHASE 2b, OPEN-LABEL STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF VACCINE CANDIDATE BNT162b2 IN IMMUNOCOMPROMISED PARTICIPANTS ≥2 YEARS OF AGE
Brief Title: Study to Evaluate Safety, Tolerability & Immunogenicity of BNT162b2 in Immunocompromised Participants ≥2 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C4591024; 2021-001290-23 (EudraCT Number)
Record Dates: First submitted 2021-05-05; First posted 2021-05-21 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: SARS-CoV-2 Infection, COVID19
Keywords: COVID19; Coronavirus; Vaccine; SARS-CoV-2; RNA Vaccine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BNT162b2 (Experimental): Intramuscular Injection
  Interventions: Biological: BNT162b2

INTERVENTIONS:
Biological: BNT162b2 — Intramuscular Injection

SUMMARY:
This is a 4 dose study with 124 participants (7 adults ,117 children). Adults are considered to be participants 18 years of age or older. Participants are going to be enrolled based on conditions that make them immunocompromised. Participants are going to be followed up for 6 months after dose 4, and each participant is projected to be on the study for approximately 15 months. This study will be conducted in the United States, Brazil, Germany and Mexico.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants who are ≥2 years of age at the time of enrollment (Visit 1).
2. Participants or participants' parent(s)/legal guardians, as age appropriate, who sign consent, and are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
3. Life expectancy ≥12 months (365 days) in the opinion of the investigator at enrollment (Visit 1).
4. Participants or participant's parent(s)/legal guardians, as age appropriate, who are able to be contacted by telephone throughout the study period.
5. Female participant of childbearing potential or male participant able to father children who is willing to use a highly effective method of contraception as outlined in this protocol for at least 28 days after the last dose of study intervention if at risk of pregnancy with her/his partner; or female participant not of childbearing potential or male participant not able to father children.
6. Participants who are immunocompromised by virtue of the following:

   * Having known non-small cell lung cancer (NSCLC) and is ≥18 years of age with at least 1 of the following:

     * Who received chemotherapy at least 2 weeks (14 days) before enrollment (or is treatment naïve), and is not expected to receive chemotherapy within at least 2 weeks (14 days) after dose administration; and/or
     * Receiving checkpoint inhibitor treatment (programmed cell death protein 1 (PD-1)/ programmed death-ligand 1 (PD-L1) inhibitor, cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitor) and has undergone at least 1 treatment cycle prior to enrollment (at Visit 1); or
     * Receiving targeted drug therapy treatment (epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), proto-oncogene tyrosine-protein kinase (ROS1), v-raf murine sarcoma viral oncogene homolog B1 (BRAF),rearranged during transfection (RET),hepatocyte growth factor receptor (MET), neurotrophic tyrosine kinase (NTRK) inhibitors) and has undergone at least 1 treatment cycle prior to enrollment (at Visit 1); or
   * Having known chronic lymphocytic leukemia (CLL) and is ≥18 years of age with at least 1 of the following:

     * Has asymptomatic disease (eg, Rai stage <3, Binet stage A or B) and is undergoing observation and does not receive any treatment for CLL; or
     * Receiving B-cell inhibitory monoclonal antibody treatment (anti-CD20) and has received at least 3 cycles prior to enrollment; and/or
     * Receives a Bruton tyrosine kinase (BTK) inhibitor, phosphoinositide 3-kinase (PI3K) inhibitor, or B-cell lymphoma-2 (BCL-2) inhibitor; or
   * Is currently undergoing maintenance hemodialysis treatment secondary to end-stage renal disease and is ≥18 years of age; or
   * Is on active immunomodulator therapy (eg, tumor necrosis factor alpha (TNFα) inhibitor, or tofacitinib or methotrexate) for an autoimmune or inflammatory disease disorder (eg, inflammatory arthritis, such as rheumatoid arthritis, psoriatic arthritis, and juvenile idiopathic arthritis, and inflammatory bowel disease, such as ulcerative colitis and Crohn's disease) at a stable* dose

     *Stable dose is defined as receiving the same dose for at least 3 months (84 days) with no changes in the 28 days prior to Visit 1; or
   * Receiving a solid organ transplant at least 3 months (84 days) prior to enrollment (Visit 1) and with no acute rejection episodes within 2 months (60 days) prior to enrollment (Visit 1), and is ≥2 to <18 years of age; or
   * Has had an autologous or allogenic bone marrow or stem cell transplant at least 6 months (182 days) prior to enrollment (Visit 1), with adequate immune reconstitution for immunization, in the investigator's opinion, and is ≥2 to <18 years of age
7. The participant or participant's parent(s)/legal guardian is capable of giving signed informed consent, and assent (as appropriate), which includes compliance with the requirements and restrictions listed in the ICD and in this protocol. The investigator, or a person designated by the investigator, will obtain written informed consent (and assent, as appropriate) from each study participant or participant's parent(s)/legal guardian before any study-specific activity is performed. All parent(s)/legal guardians should be fully informed, and participants should be informed to the fullest extent possible, about the study in language and terms they are able to understand. The investigator will retain the original copy of each participant's signed consent (and assent, as appropriate) document(s).

Exclusion Criteria:

1. Past clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID-19, or a past clinical diagnosis of multisystem inflammatory syndrome in children (MIS-C).
2. Participants with active graft-vs-host disease (GVHD), transplant rejection, or posttransplant lymphoproliferative disorder (PTLD), or participants who have had treatment for these conditions within 3 months (84 days) prior to study enrollment (Visit 1).
3. Participants <18 years of age whose weight is less than the 5th percentile of age-adjusted ideal body weight.
4. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
5. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
6. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
7. Participant who is pregnant or breastfeeding.
8. Participants who may be ineligible because of the number of phlebotomy assessments during this study, in the opinion of the investigator.
9. Participants who do not have adequate deltoid muscle mass to allow intramuscular vaccination, in the opinion of the investigator.
10. Previous vaccination with any coronavirus vaccine.
11. Ongoing, or history of, treatment with blood/plasma products or immunoglobulins within 3 months (84 days) prior to Dose 1 or planned receipt of these medications prior to Dose 4.
12. Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
13. Previous participation in other studies involving study intervention containing lipid nanoparticle (LNPs).
14. Participants who are direct descendants (child or grandchild) of investigational site staff members or Pfizer/BioNTech employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
15. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-07-23 (Actual); Study Completion 2023-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- United States (14):
  - Ochsner Clinic Foundation, Jefferson, Louisiana
  - Ochsner Medical Center - Jefferson Highway, Jefferson, Louisiana
  - Ochsner Clinic Foundation, Kenner, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Ochsner Medical Center - Jefferson Highway, New Orleans, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - Henry Ford Hospital - Research Pharmacy, Detroit, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cincinnati Children's Hospital Vaccine Research Center, Cincinnati, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Research Institute: Building Cure, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington
- Brazil (4):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - GRAACC - Grupo de Apoio ao Adolescente e à Criança com Câncer, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- Germany (7):
  - Charite - Universitaetsmedizin Berlin - Campus Virchow-Klinikum (CVK), Berlin
  - Charité - Universitaetsmedizin, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - IKF Pneumologie GmbH & Co KG, Frankfurt am Main
  - Studiengesellschaft BSF UG., Halle
  - Studiengesellschaft BSF Unternehmergesellschaft, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
- Mexico (2):
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" de la Universidad Autonoma de Nuevo Leon, Monterrey, N.L.
  - Centro Médico Zambrano Hellion, San Pedro Garza García, Nuevo León

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591024

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 124 participants were enrolled in this study.
Groups:
- (Greater Than or Equal to (>=) 2 to Less Than (<) 5 Years With Immunomodulatory Therapy: Participants aged >=2 to <5 years received immunomodulator therapy for an autoimmune inflammatory disorder were administered four doses of 3 microgram (mcg) of BNT162b2 intramuscularly. The first 2 doses were separated by 21 days, the third dose was administered 28 days after Dose 2 and fourth dose was administered 3 to 6 months after Dose 3.
- >=2 to <5 Years With Solid Organ Transplant: Participants aged >=2 to <5 years who had solid organ transplant were administered four doses of 3 mcg of BNT162b2 intramuscularly. The first 2 doses were separated by 21 days, the third dose was administered 28 days after Dose 2 and fourth dose was administered 3 to 6 months after Dose 3.
- >=2 to <5 Years With Stem Cell Transplant: Participants aged >=2 to <5 years who had stem cell transplant were administered four doses of 3 mcg of BNT162b2 intramuscularly. The first 2 doses were separated by 21 days, the third dose was administered 28 days after Dose 2 and fourth dose was administered 3 to 6 months after Dose 3.
- >=5 to <12 Years With Immunomodulatory Therapy: Participants aged >=5 to <12 years received immunomodulator therapy for an autoimmune inflammatory disorder were administered four doses of 10 mcg of BNT162b2 intramuscularly. The first 2 doses were separated by 21 days, the third dose was administered 28 days after Dose 2 and fourth dose was administered 3 to 6 months after Dose 3.
- >=5 to <12 Years With Solid Organ Transplant: Participants aged >=5 to <12 years who had solid organ transplant were administered four doses of 10 mcg of BNT162b2 intramuscularly. The first 2 doses were separated by 21 days, the third dose was administered 28 days after Dose 2 and fourth dose was administered 3 to 6 months after Dose 3.
- >=5 to <12 Years With Stem Cell Transplant: Participants aged >=5 to <12 years who had stem cell transplant were administered four doses of 10 mcg of BNT162b2 intramuscularly. The first 2 doses were separated by 21 days, the third dose was administered 28 days after Dose 2 and fourth dose was administered 3 to 6 months after Dose 3.
- >=12 to <18 Years With Immunomodulatory Therapy: Participants aged >=12 to <18 years received immunomodulator therapy for an autoimmune inflammatory disorder were administered four doses of 30 mcg of BNT162b2 intramuscularly. The first 2 doses were separated by 21 days, the third dose was administered 28 days after Dose 2 and fourth dose was administered 3 to 6 months after Dose 3.
- >=12 to <18 Years With Solid Organ Transplant: Participants aged >=12 to <18 years who had solid organ transplant were administered four doses of 30 mcg of BNT162b2 intramuscularly. The first 2 doses were separated by 21 days, the third dose was administered 28 days after Dose 2 and fourth dose was administered 3 to 6 months after Dose 3.
- >=12 to <18 Years With Stem Cell Transplant: Participants aged >=12 to <18 years who had stem cell transplant were administered four doses of 30 mcg of BNT162b2 intramuscularly. The first 2 doses were separated by 21 days, the third dose was administered 28 days after Dose 2 and fourth dose was administered 3 to 6 months after Dose 3.
- >=18 Years With Immunomodulatory Therapy: Participants aged >=18 years received immunomodulator therapy for an autoimmune inflammatory disorder were administered four doses of 30 mcg of BNT162b2 intramuscularly. The first 2 doses were separated by 21 days, the third dose was administered 28 days after Dose 2 and fourth dose was administered 3 to 6 months after Dose 3.
- >=18 Years With Non-Small Cell Lung Cancer: Participants with non-small cell lung cancer aged >=18 years were administered four doses of 30 mcg of BNT162b2 intramuscularly. The first 2 doses were separated by 21 days, the third dose was administered 28 days after Dose 2 and fourth dose was administered 3 to 6 months after Dose 3.
- >= 18 Years With Haemodialysis: Participants undergone maintenance haemodialysis treatment aged >=18 years were administered four doses of 30 mcg of BNT162b2 intramuscularly. The first 2 doses were separated by 21 days, the third dose was administered 28 days after Dose 2 and fourth dose was planned to be administered 3 to 6 months after Dose 3.
Period: Overall Study
Arm/Group | (Greater Than or Equal to (>=) 2 to Less Than (<) 5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Started | 9 | 15 | 13 | 19 | 24 | 22 | 7 | 1 | 7 | 5 | 1 | 1
Dose 1 | 9 | 15 | 13 | 19 | 24 | 22 | 7 | 1 | 7 | 5 | 1 | 1
Dose 2 | 9 | 15 | 12 | 19 | 24 | 22 | 7 | 1 | 7 | 5 | 1 | 1
Dose 3 | 9 | 15 | 11 | 17 | 24 | 22 | 7 | 1 | 6 | 5 | 1 | 1
Dose 4 | 7 | 13 | 6 | 14 | 20 | 17 | 5 | 1 | 3 | 3 | 1 | 0
Completed | 7 | 12 | 6 | 16 | 20 | 18 | 5 | 0 | 3 | 3 | 1 | 0
Not Completed | 2 | 3 | 7 | 3 | 4 | 4 | 2 | 1 | 4 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by parent/guardian | 2 | 3 | 3 | 1 | 3 | 2 | 1 | 0 | 3 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Refused further study procedures | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study intervention. To avoid risk of identification of participant, any baseline measure data is not disclosed for reporting arm including (>=18 Years with Non-Small Cell Lung Cancer, >= 18 Years with Haemodialysis) and baseline measure data other than age is not disclosed for reporting arm (>=12 to <18 Years with Solid Organ Transplant) and reported the participant under category- Not Disclosed
Groups:
- >=2 to <5 Years With Immunomodulatory Therapy: Participants aged >=2 to <5 years received immunomodulator therapy for an autoimmune inflammatory disorder were administered four doses of 3 microgram (mcg) of BNT162b2 intramuscularly. The first 2 doses were separated by 21 days, the third dose was administered 28 days after Dose 2 and fourth dose was administered 3 to 6 months after Dose 3.
- Total: Total of all reporting groups
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis | Total
Number analyzed (Participants) | 9 | 15 | 13 | 19 | 24 | 22 | 7 | 1 | 7 | 5 | 1 | 1 | 124
Age, Customized [Count of Participants; unit: Participants] — Participant in >=18 Years with Non-Small Cell Lung Cancer and >= 18 Years with Haemodialysis is not disclosed to avoid risk of identification and kept under category "Not disclosed".
  Participants
    Children (2-11 years) | 9 | 15 | 13 | 19 | 24 | 22 | 0 | 0 | 0 | 0 | 0 | 0 | 102
    Adolescents (12-17 years) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 7 | 0 | 0 | 0 | 15
    Adults (18-64 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
    From 65-84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
    Not disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Sex/Gender, Customized [Count of Participants; unit: Participants] — Participant in 12 to <18 Years with Solid Organ Transplant, >=18 Years with Non-Small Cell Lung Cancer, >= 18 Years with Haemodialysis is not disclosed to avoid risk of identification and kept under category "Not disclosed".
  Participants
    Female | 4 | 8 | 3 | 12 | 9 | 5 | 2 | 0 | 5 | 3 | 0 | 0 | 51
    Male | 5 | 7 | 10 | 7 | 15 | 17 | 5 | 0 | 2 | 2 | 0 | 0 | 70
    Not disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity is reported. Participant in 12 to <18 Years with Solid Organ Transplant, >=18 Years with Non-Small Cell Lung Cancer, >= 18 Years with Haemodialysis is not disclosed to avoid risk of identification and kept under category "Not disclosed".
  Participants
    Hispanic or Latino | 1 | 1 | 4 | 6 | 2 | 2 | 3 | 0 | 1 | 2 | 0 | 0 | 22
    Not Hispanic or Latino | 8 | 14 | 9 | 13 | 22 | 19 | 4 | 0 | 6 | 3 | 0 | 0 | 98
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Not Disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race is reported. Participant in 12 to <18 Years with Solid Organ Transplant, >=18 Years with Non-Small Cell Lung Cancer, >= 18 Years with Haemodialysis is not disclosed to avoid risk of identification and kept under category "Not disclosed".
  Participants
    Asian | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
    Black or African American | 0 | 2 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 8
    White | 9 | 11 | 12 | 17 | 21 | 19 | 6 | 0 | 7 | 1 | 0 | 0 | 103
    More than one race | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
    Unknown or Not Reported | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
    Not disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV 2) Neutralizing Titers at 1 Month After Vaccination 3 in Participants Aged >=2 to <5 Years Without Serological or Virological Evidence of Past SARS-CoV-2 Infection
Description: GMTs and corresponding 2-sided confidence intervals (CIs) were calculated by exponentiating mean logarithm of titers and corresponding CIs (based on Student's t distribution). Assay results below lower limit of quantification (LLOQ) were set to 0.5*LLOQ. Participants who had no serological or virological evidence (prior to the subsequent blood sample collection) of past SARS-CoV-2 infection (i.e, negative N-binding antibody [serum] result at any visit prior to subsequent time point, SARS-CoV-2 not detected by NAAT [nasal swab] until prior vaccination, and negative NAAT [nasal swab] result at any unscheduled visit prior to subsequent blood sample collection) and had no medical history of COVID-19 were included in the analysis. Analysis was performed in Dose 3 Evaluable Immunogenicity population (EIP).
Time Frame: 1 Month after Vaccination 3
Population: Dose 3 EIP= all participants who received 3 doses of vaccine with Dose 2 and Dose 3 within predefined window, had at least 1 valid & determinate immunogenicity result from sample collected within appropriate window (28 to 42 days, inclusive, after Dose 3); had no other important protocol deviations as determined by clinician. No participants qualified for Dose 3 EIP without prior evidence of past SARS-CoV-2 infection up to 1 month after dose 3 in '>=2 to <5 years with stem cell transplant' arm.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 5 | 6 | 0
Titers | 600.2 [77.8 to 4629.8] | 884.7 [176.7 to 4430.6] |

2. Primary Outcome: GMTs of SARS-CoV-2 Neutralizing Titers at 1 Month After Vaccination 3 in Participants Aged >=5 to <12 Years Without Serological or Virological Evidence of Past SARS-CoV-2 Infection
Description: GMTs and corresponding 2-sided CIs were calculated by exponentiating mean logarithm of titers and corresponding CIs (based on Student's t distribution). Assay results below LLOQ were set to 0.5*LLOQ. Participants who had no serological or virological evidence (prior to the subsequent blood sample collection) of past SARS-CoV-2 infection (i.e, negative N-binding antibody [serum] result at any visit prior to subsequent time point, SARS-CoV-2 not detected by NAAT [nasal swab] until prior vaccination, and negative NAAT [nasal swab] result at any unscheduled visit prior to subsequent blood sample collection) and had no medical history of COVID-19 were included in the analysis. Analysis was performed in Dose 3 EIP.
Time Frame: 1 Month after Vaccination 3
Population: Dose 3 EIP= all randomized participants who received 3 doses of vaccine with Dose 2 and Dose 3 received within the predefined window, had at least 1 valid and determinate immunogenicity result from the blood sample collected within an appropriate window (28 to 42 days, inclusive, after Dose 3), and had no other important protocol deviations as determined by the clinician.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 6 | 9 | 11
Titers | 758.4 [123.7 to 4650.4] | 741.2 [150.6 to 3647.0] | 4592.3 [1989.5 to 10600.4]

3. Primary Outcome: GMTs of SARS-CoV-2 Neutralizing Titers at 1 Month After Vaccination 3 in Participants Aged 12 to <18 Years Without Serological or Virological Evidence of Past SARS-CoV-2 Infection
Description: as for outcome 2
Time Frame: 1 Month after Vaccination 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 1 | 1 | 2
Titers | 7330.0 [NA to NA] — 95% CI could not be calculated as only one participant was analyzed. | 43.5 [NA to NA] — 95% CI could not be calculated as only one participant was analyzed. | 2368.1 [1679.9 to 3338.3]

4. Primary Outcome: GMTs of SARS-CoV-2 Neutralizing Titers at 1 Month After Vaccination 3 in Participants Aged >=18 Years Without Serological or Virological Evidence of Past SARS-CoV-2 Infection
Description: as for outcome 2
Time Frame: 1 Month after Vaccination 3
Population: Dose 3 EIP= all participants who received 3 doses of vaccine with Dose 2 and Dose 3 within predefined window, had at least 1 valid & determinate immunogenicity result from sample collected within appropriate window (28 to 42 days, inclusive, after Dose 3); had no other important protocol deviations as determined by clinician. No participants qualified for Dose 3 EIP without prior evidence of past SARS-CoV-2 infection up to 1 month after dose 3 in '>=18 years with non small cell lung cancer' arm.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 2 | 0 | 1
Titers | 596.5 [0.1 to 3699753.4] |  | 115.0 [NA to NA] — 95% CI could not be calculated as only one participant was analyzed.

5. Primary Outcome: GMTs of SARS-CoV-2 Neutralizing Titers at 1 Month After Vaccination 4 in Participants Aged >=2 to <5 Years Without Serological or Virological Evidence of Past SARS-CoV-2 Infection
Description: GMTs and corresponding 2-sided CIs were calculated by exponentiating mean logarithm of titers and corresponding CIs (based on Student's t distribution). Assay results below LLOQ were set to 0.5*LLOQ. Participants who had no serological or virological evidence (prior to the subsequent blood sample collection) of past SARS-CoV-2 infection (i.e, negative N-binding antibody [serum] result at any visit prior to subsequent time point, SARS-CoV-2 not detected by NAAT [nasal swab] until prior vaccination, and negative NAAT [nasal swab] result at any unscheduled visit prior to subsequent blood sample collection) and had no medical history of COVID-19 were included in the analysis. Analysis was performed in Dose 4 EIP.
Time Frame: 1 Month after Vaccination 4
Population: Dose 4 EIP= all participants who received 4 doses of vaccine with Dose 2,3&4 within predefined window,had at least 1 valid & determinate immunogenicity result from sample collected within appropriate window (28 to 42 days, inclusive, after Dose 4); had no other important protocol deviations as determined by clinician. No participants qualified for Dose 4 EIP without prior evidence of past SARS-CoV-2 infection up to 1 month after dose 4 in '>=2 to <5 years with stem cell transplant' arm.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 3 | 2 | 0
Titers | 837.5 [1.4 to 518774.5] | 9576.3 [0.0 to 2070132632.7] |

6. Primary Outcome: GMTs of SARS-CoV-2 Neutralizing Titers at 1 Month After Vaccination 4 in Participants Aged >=5 to <12 Years Without Serological or Virological Evidence of Past SARS-CoV-2 Infection
Description: as for outcome 5
Time Frame: 1 Month after Vaccination 4
Population: Dose 4 EIP= all randomized participants who received 4 doses of vaccine with Dose 2, Dose 3 and Dose 4 received within the predefined window, had at least 1 valid and determinate immunogenicity result from the blood sample collected within an appropriate window (28 to 42 days, inclusive, after Dose 4), and had no other important protocol deviations as determined by the clinician.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 2 | 4 | 2
Titers | 754.2 [0.0 to 351878145.2] | 5335.3 [517.0 to 55061.8] | 5330.8 [0.0 to 113927797661576]

7. Primary Outcome: GMTs of SARS-CoV-2 Neutralizing Titers at 1 Month After Vaccination 4 in Participants Aged 12 to <18 Years Without Serological or Virological Evidence of Past SARS-CoV-2 Infection
Description: as for outcome 5
Time Frame: 1 Month after Vaccination 4
Population: Dose 4 EIP=all participants who received 4 doses of vaccine with Dose 2,3&4 within predefined window,had atleast 1 valid&determinate immunogenicity result from sample collected within appropriate window(28-42 days,inclusive,after Dose4);had no other important protocol deviations as determined by clinician.No participants qualified for Dose 4 EIP without prior evidence of past SARS-CoV-2 infection up to 1 month after dose4 in'12 to <18 years with immunomodulatory therapy&stem cell transplant'arm.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 0 | 1 | 0
Titers |  | 2845.0 [NA to NA] — 95% CI could not be calculated as only one participant was analyzed. |

8. Primary Outcome: GMTs of SARS-CoV-2 Neutralizing Titers at 1 Month After Vaccination 4 in Participants Aged >=18 Years Without Serological or Virological Evidence of Past SARS-CoV-2 Infection
Description: GMTs and corresponding 2-sided CIs were calculated by exponentiating mean logarithm of titers and corresponding CIs (based on Student's t distribution). Assay results below lower limit of quantification (LLOQ) were set to 0.5*LLOQ. Participants who had no serological or virological evidence (prior to the subsequent blood sample collection) of past SARS-CoV-2 infection (i.e, negative N-binding antibody [serum] result at any visit prior to subsequent time point, SARS-CoV-2 not detected by NAAT [nasal swab] until prior vaccination, and negative NAAT [nasal swab] result at any unscheduled visit prior to subsequent blood sample collection) and had no medical history of COVID-19 were included in the analysis. Analysis was performed in Dose 4 EIP .
Time Frame: 1 Month after Vaccination 4
Population: Dose 4 EIP=all participants who received 4 doses of vaccine with Dose 2,3&4 within predefined window,had at least 1 valid& determinate immunogenicity result from sample collected within appropriate window (28 to 42 days, inclusive, after Dose 4); had no other important protocol deviations as determined by clinician. No participants qualified for Dose 4 EIP without prior evidence of past SARS-CoV-2 infection up to 1 month after dose 4 in '>=18 years with non-small cell lung cancer&hemodialysis'
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 1 | 0 | 0
Titers | 1474.0 [NA to NA] — 95% CI could not be calculated as only one participant was analyzed. |  |

9. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 1 in Participants Aged >=2 to <5 Years
Description: Local reactions were collected in an electronic diary (e-diary) or during unscheduled clinical assessments from Day 1 to 7 after vaccination 1. Redness and swelling were measured and recorded in measuring device units (mdu) where, 1 mdu =0.5 centimeter (cm) and were graded as mild (>0.5 to 2.0 cm), moderate (>2.0 to 7.0 cm), severe (>7.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (emergency room [ER] visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Reactions reported as adverse events in case report form within 7 days of study vaccination were also included. Two-sided 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 1
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 9 | 15 | 13
Percentage of participants
  Redness: Any | 11.1 (0.3) [0.3 to 48.2] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 24.7]
  Redness: Mild | 11.1 (0.3) [0.3 to 48.2] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 24.7]
  Redness: Moderate | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Redness: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Redness: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Swelling: Any | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Swelling: Mild | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Swelling: Moderate | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Swelling: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Swelling: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Pain at the injection site: Any | 11.1 (0.3) [0.3 to 48.2] | 13.3 (1.7) [1.7 to 40.5] | 23.1 (5.0) [5.0 to 53.8]
  Pain at the injection site: Mild | 11.1 (0.3) [0.3 to 48.2] | 13.3 (1.7) [1.7 to 40.5] | 23.1 (5.0) [5.0 to 53.8]
  Pain at the injection site: Moderate | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Pain at the injection site: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Pain at the injection site: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]

10. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 1 in Participants Aged >=5 to <12 Years
Description: Local reactions were collected in e-diary or during unscheduled clinical assessments from Day 1 to Day 7 after vaccination 1.Redness and swelling were measured and recorded in mdu where, 1 mdu =0.5 cm and were graded as mild (>0.5 to 2.0 cm),moderate (>2.0 to 7.0 cm), severe (>7.0 cm) and Grade 4(necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 ER visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Reactions reported as adverse events in case report form within 7 days of study vaccination were also included. Two-sided 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 1
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 19 | 24 | 22
Percentage of participants
  Redness: Any | 10.5 (1.3) [1.3 to 33.1] | 8.3 (1.0) [1.0 to 27.0] | 9.1 (1.1) [1.1 to 29.2]
  Redness: Mild | 10.5 (1.3) [1.3 to 33.1] | 4.2 (0.1) [0.1 to 21.1] | 4.5 (0.1) [0.1 to 22.8]
  Redness: Moderate | 0 (0.0) [0.0 to 17.6] | 4.2 (0.1) [0.1 to 21.1] | 4.5 (0.1) [0.1 to 22.8]
  Redness: Severe | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Redness: Grade 4 | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Swelling: Any | 5.3 (0.1) [0.1 to 26.0] | 4.2 (0.1) [0.1 to 21.1] | 18.2 (5.2) [5.2 to 40.3]
  Swelling: Mild | 5.3 (0.1) [0.1 to 26.0] | 0 (0.0) [0.0 to 14.2] | 13.6 (2.9) [2.9 to 34.9]
  Swelling: Moderate | 0 (0.0) [0.0 to 17.6] | 4.2 (0.1) [0.1 to 21.1] | 4.5 (0.1) [0.1 to 22.8]
  Swelling: Severe | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Swelling: Grade 4 | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Pain at the injection site: Any | 73.7 (48.8) [48.8 to 90.9] | 58.3 (36.6) [36.6 to 77.9] | 54.5 (32.2) [32.2 to 75.6]
  Pain at the injection site: Mild | 52.6 (28.9) [28.9 to 75.6] | 50.0 (29.1) [29.1 to 70.9] | 45.5 (24.4) [24.4 to 67.8]
  Pain at the injection site: Moderate | 21.1 (6.1) [6.1 to 45.6] | 8.3 (1.0) [1.0 to 27.0] | 9.1 (1.1) [1.1 to 29.2]
  Pain at the injection site: Severe | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Pain at the injection site: Grade 4 | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]

11. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 1 in Participants Aged >=12 to <18 Years
Description: Local reactions were collected in e-diary or during unscheduled clinical assessments from Day 1 to Day 7 after vaccination 1. Redness and swelling were measured and recorded in mdu where, 1 mdu =0.5 cm and were graded as mild (> 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (ER visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Reactions reported as adverse events in case report form within 7 days of study vaccination were also included. Two-sided 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 1
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 7 | 1 | 7
Percentage of participants
  Redness: Any | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 97.5] | 14.3 (0.4) [0.4 to 57.9]
  Redness: Mild | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 97.5] | 14.3 (0.4) [0.4 to 57.9]
  Redness: Moderate | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Redness: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Redness: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Swelling: Any | 28.6 (3.7) [3.7 to 71.0] | 100.0 (2.5) [2.5 to 100.0] | 14.3 (0.4) [0.4 to 57.9]
  Swelling: Mild | 0 (0.0) [0.0 to 41.0] | 100.0 (2.5) [2.5 to 100.0] | 0 (0.0) [0.0 to 41.0]
  Swelling: Moderate | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 97.5] | 14.3 (0.4) [0.4 to 57.9]
  Swelling: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Swelling: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Pain at the injection site: Any | 85.7 (42.1) [42.1 to 99.6] | 100.0 (2.5) [2.5 to 100.0] | 57.1 (18.4) [18.4 to 90.1]
  Pain at the injection site: Mild | 71.4 (29.0) [29.0 to 96.3] | 100.0 (2.5) [2.5 to 100.0] | 28.6 (3.7) [3.7 to 71.0]
  Pain at the injection site: Moderate | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 28.6 (3.7) [3.7 to 71.0]
  Pain at the injection site: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Pain at the injection site: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]

12. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 1 in Participants Aged >=18 Years
Description: Local reactions were collected in e-diary or during unscheduled clinical assessments from Day 1 to Day 7 after vaccination 1. Redness and swelling were measured and recorded in mdu where, 1 mdu =0.5 cm and were graded as mild (> 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (ER visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Reactions reported as adverse events in case report form within 7 days of study vaccination also included. Two-sided 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 1
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 5 | 1 | 1
Percentage of participants
  Redness: Any | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Redness: Mild | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Redness: Moderate | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Redness: Severe | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Redness: Grade 4 | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Swelling: Any | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Swelling: Mild | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Swelling: Moderate | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Swelling: Severe | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Swelling: Grade 4 | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Pain at injection site: Any | 80.0 (28.4) [28.4 to 99.5] | 100.0 (2.5) [2.5 to 100.0] | 100.0 (2.5) [2.5 to 100.0]
  Pain at injection site: Mild | 40.0 (5.3) [5.3 to 85.3] | 100.0 (2.5) [2.5 to 100.0] | 0 (0.0) [0.0 to 97.5]
  Pain at injection site: Moderate | 40.0 (5.3) [5.3 to 85.3] | 0 (0.0) [0.0 to 97.5] | 100.0 (2.5) [2.5 to 100.0]
  Pain at injection site: Severe | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Pain at injection site: Grade 4 | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]

13. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 2 in Participants Aged >=2 to <5 Years
Description: Local reactions collected in e-diary or during unscheduled clinical assessments from Day 1 to Day 7 after vaccination 2. Redness and swelling were measured and recorded in mdu where, 1 mdu =0.5 cm and were graded as mild (>0.5 to 2.0 cm),moderate(>2.0 to 7.0 cm), severe(>7.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis[redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate(interfered with activity), severe(prevented daily activity),Grade 4(ER visit or hospitalization for severe pain at injection site).Grade 4 were classified by investigator or medically qualified person. Reactions reported as adverse events in case report form within 7 days of study vaccination were also included. Two-sided 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 2
Population: Safety population consisted of all participants who received at least 1 dose of study intervention. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 9 | 15 | 11
Percentage of participants
  Redness: Any: number analyzed (Participants) | 9 | 15 | 10
  Redness: Any | 0 [0.0 to 33.6] | 6.7 [0.2 to 31.9] | 0 [0.0 to 30.8]
  Redness: Mild: number analyzed (Participants) | 9 | 15 | 10
  Redness: Mild | 0 [0.0 to 33.6] | 6.7 [0.2 to 31.9] | 0 [0.0 to 30.8]
  Redness: Moderate: number analyzed (Participants) | 9 | 15 | 10
  Redness: Moderate | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Redness: Severe: number analyzed (Participants) | 9 | 15 | 10
  Redness: Severe | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Redness: Grade 4: number analyzed (Participants) | 9 | 15 | 10
  Redness: Grade 4 | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Swelling: Any: number analyzed (Participants) | 9 | 15 | 10
  Swelling: Any | 0 [0.0 to 33.6] | 6.7 [0.2 to 31.9] | 0 [0.0 to 30.8]
  Swelling: Mild: number analyzed (Participants) | 9 | 15 | 10
  Swelling: Mild | 0 [0.0 to 33.6] | 6.7 [0.2 to 31.9] | 0 [0.0 to 30.8]
  Swelling: Moderate: number analyzed (Participants) | 9 | 15 | 10
  Swelling: Moderate | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Swelling: Severe: number analyzed (Participants) | 9 | 15 | 10
  Swelling: Severe | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Swelling: Grade 4: number analyzed (Participants) | 9 | 15 | 10
  Swelling: Grade 4 | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Pain at injection site: Any | 11.1 [0.3 to 48.2] | 20.0 [4.3 to 48.1] | 9.1 [0.2 to 41.3]
  Pain at injection site: Mild | 11.1 [0.3 to 48.2] | 20.0 [4.3 to 48.1] | 9.1 [0.2 to 41.3]
  Pain at injection site: Moderate | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 28.5]
  Pain at injection site: Severe | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 28.5]
  Pain at injection site: Grade 4 | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 28.5]

14. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 2 in Participants Aged >=5 to <12 Years
Description: Local reactions were collected in e-diary or during unscheduled clinical assessments from Day 1 to Day 7 after vaccination 2.Redness and swelling were measured and recorded in mdu where, 1 mdu =0.5 cm and were graded as mild (>0.5 to 2.0 cm),moderate (>2.0 to 7.0 cm), severe (>7.0 cm) and Grade 4(necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 ER visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Reactions reported as adverse events in case report form within 7 days of study vaccination were also included. Two-sided 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 2
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 19 | 24 | 22
Percentage of participants
  Redness: Any | 10.5 (1.3) [1.3 to 33.1] | 12.5 (2.7) [2.7 to 32.4] | 22.7 (7.8) [7.8 to 45.4]
  Redness: Mild | 10.5 (1.3) [1.3 to 33.1] | 4.2 (0.1) [0.1 to 21.1] | 13.6 (2.9) [2.9 to 34.9]
  Redness: Moderate | 0 (0.0) [0.0 to 17.6] | 8.3 (1.0) [1.0 to 27.0] | 9.1 (1.1) [1.1 to 29.2]
  Redness: Severe | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Redness: Grade 4 | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Swelling: Any | 10.5 (1.3) [1.3 to 33.1] | 8.3 (1.0) [1.0 to 27.0] | 31.8 (13.9) [13.9 to 54.9]
  Swelling: Mild | 10.5 (1.3) [1.3 to 33.1] | 4.2 (0.1) [0.1 to 21.1] | 9.1 (1.1) [1.1 to 29.2]
  Swelling: Moderate | 0 (0.0) [0.0 to 17.6] | 4.2 (0.1) [0.1 to 21.1] | 22.7 (7.8) [7.8 to 45.4]
  Swelling: Severe | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Swelling: Grade 4 | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Pain at injection site: Any | 68.4 (43.4) [43.4 to 87.4] | 62.5 (40.6) [40.6 to 81.2] | 50.0 (28.2) [28.2 to 71.8]
  Pain at injection site: Mild | 52.6 (28.9) [28.9 to 75.6] | 45.8 (25.6) [25.6 to 67.2] | 22.7 (7.8) [7.8 to 45.4]
  Pain at injection site: Moderate | 15.8 (3.4) [3.4 to 39.6] | 16.7 (4.7) [4.7 to 37.4] | 27.3 (10.7) [10.7 to 50.2]
  Pain at injection site: Severe | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Pain at injection site: Grade 4 | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]

15. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 2 in Participants Aged >=12 to <18 Years
Description: Local reactions were collected in e-diary or during unscheduled clinical assessments from Day 1 to Day 7 after vaccination 2. Redness and swelling were measured and recorded in mdu where, 1 mdu =0.5 cm and were graded as mild (> 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (ER visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Reactions reported as adverse events in case report form within 7 days of study vaccination were also included. Two-sided 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 2
Population: Safety population consisted of all participants who received at least 1 dose of study intervention. 'Number Analyzed (n)' signifies participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 7 | 1 | 7
Percentage of participants
  Redness: Any: number analyzed (Participants) | 7 | 1 | 6
  Redness: Any | 14.3 [0.4 to 57.9] | 0 [0.0 to 97.5] | 16.7 [0.4 to 64.1]
  Redness: Mild: number analyzed (Participants) | 7 | 1 | 6
  Redness: Mild | 14.3 [0.4 to 57.9] | 0 [0.0 to 97.5] | 16.7 [0.4 to 64.1]
  Redness: Moderate: number analyzed (Participants) | 7 | 1 | 6
  Redness: Moderate | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Redness: Severe: number analyzed (Participants) | 7 | 1 | 6
  Redness: Severe | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Redness: Grade 4: number analyzed (Participants) | 7 | 1 | 6
  Redness: Grade 4 | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Swelling: Any: number analyzed (Participants) | 7 | 1 | 6
  Swelling: Any | 28.6 [3.7 to 71.0] | 0 [0.0 to 97.5] | 16.7 [0.4 to 64.1]
  Swelling: Mild: number analyzed (Participants) | 7 | 1 | 6
  Swelling: Mild | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 16.7 [0.4 to 64.1]
  Swelling: Moderate: number analyzed (Participants) | 7 | 1 | 6
  Swelling: Moderate | 28.6 [3.7 to 71.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Swelling: Severe: number analyzed (Participants) | 7 | 1 | 6
  Swelling: Severe | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Swelling: Grade 4: number analyzed (Participants) | 7 | 1 | 6
  Swelling: Grade 4 | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Pain at injection site: Any | 85.7 [42.1 to 99.6] | 100.0 [2.5 to 100.0] | 57.1 [18.4 to 90.1]
  Pain at injection site: Mild | 57.1 [18.4 to 90.1] | 100.0 [2.5 to 100.0] | 28.6 [3.7 to 71.0]
  Pain at injection site: Moderate | 28.6 [3.7 to 71.0] | 0 [0.0 to 97.5] | 28.6 [3.7 to 71.0]
  Pain at injection site: Severe | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 41.0]
  Pain at injection site: Grade 4 | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 41.0]

16. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 2 in Participants Aged >=18 Years
Description: as for outcome 15
Time Frame: Day 1 to Day 7 after Vaccination 2
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 5 | 1 | 1
Percentage of participants
  Redness: Any | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Redness: Mild | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Redness: Moderate | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Redness: Severe | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Redness: Grade 4 | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Swelling: Any | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Swelling: Mild | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Swelling: Moderate | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Swelling: Severe | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Swelling: Grade 4 | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Pain at injection site: Any | 80.0 (28.4) [28.4 to 99.5] | 100.0 (2.5) [2.5 to 100.0] | 0 (0.0) [0.0 to 97.5]
  Pain at injection site: Mild | 60.0 (14.7) [14.7 to 94.7] | 100.0 (2.5) [2.5 to 100.0] | 0 (0.0) [0.0 to 97.5]
  Pain at injection site: Moderate | 20.0 (0.5) [0.5 to 71.6] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Pain at injection site: Severe | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Pain at injection site: Grade 4 | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]

17. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 3 in Participants Aged >=2 to <5 Years
Description: Local reactions were collected in e-diary or during unscheduled clinical assessments from Day 1 to Day 7 after vaccination 3.Redness and swelling were measured and recorded in mdu where, 1 mdu =0.5 cm and were graded as mild (>0.5 to 2.0 cm),moderate (>2.0 to 7.0 cm), severe (>7.0 cm) and Grade 4(necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 ER visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Reactions reported as adverse events in case report form within 7 days of study vaccination were also included. Two-sided 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 3
Population: Safety population consisted of all participants who received at least 1 dose of study intervention. Here, 'Overall Number of Participants Analyzed (N)' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 9 | 15 | 11
Percentage of participants
  Redness: Any | 11.1 (0.3) [0.3 to 48.2] | 13.3 (1.7) [1.7 to 40.5] | 0 (0.0) [0.0 to 28.5]
  Redness: Mild | 0 (0.0) [0.0 to 33.6] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 28.5]
  Redness: Moderate | 11.1 (0.3) [0.3 to 48.2] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 28.5]
  Redness: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Redness: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Swelling: Any | 11.1 (0.3) [0.3 to 48.2] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 28.5]
  Swelling: Mild | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Swelling: Moderate | 11.1 (0.3) [0.3 to 48.2] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 28.5]
  Swelling: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Swelling: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Pain at injection site: Any | 22.2 (2.8) [2.8 to 60.0] | 13.3 (1.7) [1.7 to 40.5] | 9.1 (0.2) [0.2 to 41.3]
  Pain at injection site: Mild | 0 (0.0) [0.0 to 33.6] | 13.3 (1.7) [1.7 to 40.5] | 9.1 (0.2) [0.2 to 41.3]
  Pain at injection site: Moderate | 22.2 (2.8) [2.8 to 60.0] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Pain at injection site: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Pain at injection site: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]

18. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 3 in Participants Aged >=5 to <12 Years
Description: as for outcome 17
Time Frame: Day 1 to Day 7 after Vaccination 3
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 17 | 23 | 21
Percentage of participants
  Redness: Any | 29.4 (10.3) [10.3 to 56.0] | 4.3 (0.1) [0.1 to 21.9] | 14.3 (3.0) [3.0 to 36.3]
  Redness: Mild | 17.6 (3.8) [3.8 to 43.4] | 0 (0.0) [0.0 to 14.8] | 9.5 (1.2) [1.2 to 30.4]
  Redness: Moderate | 11.8 (1.5) [1.5 to 36.4] | 4.3 (0.1) [0.1 to 21.9] | 4.8 (0.1) [0.1 to 23.8]
  Redness: Severe | 0 (0.0) [0.0 to 19.5] | 0 (0.0) [0.0 to 14.8] | 0 (0.0) [0.0 to 16.1]
  Redness: Grade 4 | 0 (0.0) [0.0 to 19.5] | 0 (0.0) [0.0 to 14.8] | 0 (0.0) [0.0 to 16.1]
  Swelling: Any | 17.6 (3.8) [3.8 to 43.4] | 8.7 (1.1) [1.1 to 28.0] | 14.3 (3.0) [3.0 to 36.3]
  Swelling: Mild | 5.9 (0.1) [0.1 to 28.7] | 0 (0.0) [0.0 to 14.8] | 9.5 (1.2) [1.2 to 30.4]
  Swelling: Moderate | 11.8 (1.5) [1.5 to 36.4] | 8.7 (1.1) [1.1 to 28.0] | 4.8 (0.1) [0.1 to 23.8]
  Swelling: Severe | 0 (0.0) [0.0 to 19.5] | 0 (0.0) [0.0 to 14.8] | 0 (0.0) [0.0 to 16.1]
  Swelling: Grade 4 | 0 (0.0) [0.0 to 19.5] | 0 (0.0) [0.0 to 14.8] | 0 (0.0) [0.0 to 16.1]
  Pain at injection site: Any | 70.6 (44.0) [44.0 to 89.7] | 26.1 (10.2) [10.2 to 48.4] | 57.1 (34.0) [34.0 to 78.2]
  Pain at injection site: Mild | 35.3 (14.2) [14.2 to 61.7] | 21.7 (7.5) [7.5 to 43.7] | 42.9 (21.8) [21.8 to 66.0]
  Pain at injection site: Moderate | 35.3 (14.2) [14.2 to 61.7] | 4.3 (0.1) [0.1 to 21.9] | 14.3 (3.0) [3.0 to 36.3]
  Pain at injection site: Severe | 0 (0.0) [0.0 to 19.5] | 0 (0.0) [0.0 to 14.8] | 0 (0.0) [0.0 to 16.1]
  Pain at injection site: Grade 4 | 0 (0.0) [0.0 to 19.5] | 0 (0.0) [0.0 to 14.8] | 0 (0.0) [0.0 to 16.1]

19. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 3 in Participants Aged >=12 to <18 Years
Description: Local reactions were collected in e-diary or during unscheduled clinical assessments from Day 1 to Day 7 after vaccination 3. Redness and swelling were measured and recorded in mdu where, 1 mdu =0.5 cm and were graded as mild >2.0 to 5.0 cm), moderate(>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate(interfered with activity), severe(prevented daily activity) and Grade 4(ER visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Reactions reported as adverse events in case report form within 7 days of study vaccination were also included. Two-sided 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 3
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 7 | 1 | 6
Percentage of participants
  Redness: Any | 14.3 [0.4 to 57.9] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Redness: Mild | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Redness: Moderate | 14.3 [0.4 to 57.9] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Redness: Severe | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Redness: Grade 4 | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Swelling: Any | 28.6 [3.7 to 71.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Swelling: Mild | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Swelling: Moderate | 28.6 [3.7 to 71.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Swelling: Severe | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Swelling: Grade 4 | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Pain at injection site: Any | 71.4 [29.0 to 96.3] | 100.0 [2.5 to 100.0] | 66.7 [22.3 to 95.7]
  Pain at injection site: Mild | 28.6 [3.7 to 71.0] | 100.0 [2.5 to 100.0] | 33.3 [4.3 to 77.7]
  Pain at injection site: Moderate | 42.9 [9.9 to 81.6] | 0 [0.0 to 97.5] | 33.3 [4.3 to 77.7]
  Pain at injection site: Severe | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Pain at injection site: Grade 4 | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]

20. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 3 in Participants Aged >=18 Years
Description: Local reactions were collected in e-diary or during unscheduled clinical assessments from Day 1 to Day 7 after vaccination 3. Redness and swelling were measured and recorded in mdu where, 1 mdu =0.5 cm and were graded as mild (> 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (ER visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Reactions reported as adverse events in case report form within 7 days of study vaccination were also included. Two-sided 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 3
Population: Safety population consisted of all participants who received at least 1 dose of study intervention. Here, 'Overall Number of Participants Analyzed (N)' signifies participants evaluable for this outcome measure. Data is not reported for ">=18 Years with Non-Small Cell Lung Cancer" arm as e-diary data is not transmitted (i.e. participants had not reported the data for the entire e- diary collection period).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 4 | 0 | 1
Percentage of participants
  Redness: Any | 25.0 (0.6) [0.6 to 80.6] |  | 0 (0.0) [0.0 to 97.5]
  Redness: Mild | 25.0 (0.6) [0.6 to 80.6] |  | 0 (0.0) [0.0 to 97.5]
  Redness: Moderate | 0 (0.0) [0.0 to 60.2] |  | 0 (0.0) [0.0 to 97.5]
  Redness: Severe | 0 (0.0) [0.0 to 60.2] |  | 0 (0.0) [0.0 to 97.5]
  Redness: Grade 4 | 0 (0.0) [0.0 to 60.2] |  | 0 (0.0) [0.0 to 97.5]
  Swelling: Any | 25.0 (0.6) [0.6 to 80.6] |  | 0 (0.0) [0.0 to 97.5]
  Swelling: Mild | 25.0 (0.6) [0.6 to 80.6] |  | 0 (0.0) [0.0 to 97.5]
  Swelling: Moderate | 0 (0.0) [0.0 to 60.2] |  | 0 (0.0) [0.0 to 97.5]
  Swelling: Severe | 0 (0.0) [0.0 to 60.2] |  | 0 (0.0) [0.0 to 97.5]
  Swelling: Grade 4 | 0 (0.0) [0.0 to 60.2] |  | 0 (0.0) [0.0 to 97.5]
  Pain at injection site: Any | 75.0 (19.4) [19.4 to 99.4] |  | 0 (0.0) [0.0 to 97.5]
  Pain at injection site: Mild | 50.0 (6.8) [6.8 to 93.2] |  | 0 (0.0) [0.0 to 97.5]
  Pain at injection site: Moderate | 25.0 (0.6) [0.6 to 80.6] |  | 0 (0.0) [0.0 to 97.5]
  Pain at injection site: Severe | 0 (0.0) [0.0 to 60.2] |  | 0 (0.0) [0.0 to 97.5]
  Pain at injection site: Grade 4 | 0 (0.0) [0.0 to 60.2] |  | 0 (0.0) [0.0 to 97.5]

21. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 4 in Participants Aged >=2 to <5 Years
Description: Local reactions were collected in e-diary or during unscheduled clinical assessments from Day 1 to Day 7 after vaccination 4.Redness and swelling were measured and recorded in mdu where, 1 mdu =0.5 cm and were graded as mild (>0.5 to 2.0 cm),moderate (>2.0 to 7.0 cm), severe (>7.0 cm) and Grade 4(necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 ER visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Reactions reported as adverse events in case report form within 7 days of study vaccination were also included. Two-sided 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 4
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 7 | 6 | 6
Percentage of participants
  Redness: Any | 28.6 (3.7) [3.7 to 71.0] | 16.7 (0.4) [0.4 to 64.1] | 0 (0.0) [0.0 to 45.9]
  Redness: Mild | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Redness: Moderate | 14.3 (0.4) [0.4 to 57.9] | 16.7 (0.4) [0.4 to 64.1] | 0 (0.0) [0.0 to 45.9]
  Redness: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Redness: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Swelling: Any | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 45.9] | 16.7 (0.4) [0.4 to 64.1]
  Swelling: Mild | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 16.7 (0.4) [0.4 to 64.1]
  Swelling: Moderate | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Swelling: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Swelling: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Pain at injection site: Any | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 45.9] | 16.7 (0.4) [0.4 to 64.1]
  Pain at injection site: Mild | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 45.9] | 16.7 (0.4) [0.4 to 64.1]
  Pain at injection site: Moderate | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Pain at injection site: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Pain at injection site: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]

22. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 4 in Participants Aged >=5 to <12 Years
Description: as for outcome 21
Time Frame: Day 1 to Day 7 after Vaccination 4
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 12 | 19 | 15
Percentage of participants
  Redness: Any | 8.3 (0.2) [0.2 to 38.5] | 5.3 (0.1) [0.1 to 26.0] | 20.0 (4.3) [4.3 to 48.1]
  Redness: Mild | 8.3 (0.2) [0.2 to 38.5] | 5.3 (0.1) [0.1 to 26.0] | 6.7 (0.2) [0.2 to 31.9]
  Redness: Moderate | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 13.3 (1.7) [1.7 to 40.5]
  Redness: Severe | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Redness: Grade 4 | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Swelling: Any | 16.7 (2.1) [2.1 to 48.4] | 5.3 (0.1) [0.1 to 26.0] | 20.0 (4.3) [4.3 to 48.1]
  Swelling: Mild | 8.3 (0.2) [0.2 to 38.5] | 5.3 (0.1) [0.1 to 26.0] | 13.3 (1.7) [1.7 to 40.5]
  Swelling: Moderate | 8.3 (0.2) [0.2 to 38.5] | 0 (0.0) [0.0 to 17.6] | 6.7 (0.2) [0.2 to 31.9]
  Swelling: Severe | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Swelling: Grade 4 | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Pain at injection site: Any | 91.7 (61.5) [61.5 to 99.8] | 42.1 (20.3) [20.3 to 66.5] | 40.0 (16.3) [16.3 to 67.7]
  Pain at injection site: Mild | 41.7 (15.2) [15.2 to 72.3] | 31.6 (12.6) [12.6 to 56.6] | 26.7 (7.8) [7.8 to 55.1]
  Pain at injection site: Moderate | 50.0 (21.1) [21.1 to 78.9] | 10.5 (1.3) [1.3 to 33.1] | 13.3 (1.7) [1.7 to 40.5]
  Pain at injection site: Severe | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Pain at injection site: Grade 4 | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]

23. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 4 in Participants Aged >=12 to <18 Years
Description: Local reactions were collected in e-diary or during unscheduled clinical assessments from Day 1 to Day 7 after vaccination 4. Redness and swelling were measured and recorded in mdu where, 1 mdu =0.5 cm and were graded as mild (> 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (ER visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Reactions reported as adverse events in case report form within 7 days of study vaccination also included. Two-sided 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 4
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.Here, 'Overall Number of Participants Analyzed (N)' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 4 | 1 | 3
Percentage of participants
  Redness: Any | 75.0 [19.4 to 99.4] | 0 [0.0 to 97.5] | 66.7 [9.4 to 99.2]
  Redness: Mild | 75.0 [19.4 to 99.4] | 0 [0.0 to 97.5] | 66.7 [9.4 to 99.2]
  Redness: Moderate | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Redness: Severe | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Redness: Grade 4 | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Swelling: Any | 50.0 [6.8 to 93.2] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Swelling: Mild | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Swelling: Moderate | 50.0 [6.8 to 93.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Swelling: Severe | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Swelling: Grade 4 | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Pain at injection site: Any | 75.0 [19.4 to 99.4] | 100.0 [2.5 to 100.0] | 33.3 [0.8 to 90.6]
  Pain at injection site: Mild | 25.0 [0.6 to 80.6] | 100.0 [2.5 to 100.0] | 0 [0.0 to 70.8]
  Pain at injection site: Moderate | 50.0 [6.8 to 93.2] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Pain at injection site: Severe | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Pain at injection site: Grade 4 | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]

24. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 4 in Participants Aged >=18 Years
Description: Local reactions were collected in e-diary or during unscheduled clinical assessments from Day 1 to Day 7 after vaccination 4. Redness and swelling were measured and recorded in mdu where, 1 mdu =0.5 cm and were graded as mild (> 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (ER visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Reactions reported as adverse events in case report form within 7 days of study vaccination were also included. Two-sided 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 4
Population: Safety population consisted of all participants who received at least 1 dose of study intervention. Here, 'Overall Number of Participants Analyzed (N)' signifies participants evaluable for this outcome measure. Participants of >=18 years haemodialysis: group did not receive Vaccination 4 and therefore were not analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 3 | 1 | 0
Percentage of participants
  Redness: Any | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  Redness: Mild | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  Redness: Moderate | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Redness: Severe | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Redness: Grade 4 | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Swelling: Any | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  Swelling: Mild | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  Swelling: Moderate | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Swelling: Severe | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Swelling: Grade 4 | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Pain at injection site: Any | 66.7 (9.4) [9.4 to 99.2] | 100.0 (2.5) [2.5 to 100.0] |
  Pain at injection site: Mild | 33.3 (0.8) [0.8 to 90.6] | 100.0 (2.5) [2.5 to 100.0] |
  Pain at injection site: Moderate | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  Pain at injection site: Severe | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Pain at injection site: Grade 4 | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |

25. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 1 in Participants Aged >=2 to <5 Years
Description: Systemic events were recorded in an e-diary and at unscheduled clinical assessments from Day 1 to 7 after vaccination 1. Fever was defined as oral temperature >=38.0 degree C (deg C); categorized as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain: mild (did not interfere with activity), moderate (some interference with activity), severe (prevented daily routine activity).Vomiting: mild: 1-2 times in 24 hours, moderate: >2 times in 24 hours, severe: required intravenous hydration. Diarrhea: mild: 2-3 loose stools in 24 hours, moderate: 4-5 loose stools in 24 hours, severe: 6 or more loose stools in 24 hours. Grade 4 for all events: ER visit/hospitalization and were classified by investigator or medically qualified person. Events reported as AEs in the CRF within 7 days after vaccination were also included. Exact 95% CI based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 1
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 9 | 15 | 13
Percentage of participants
  Fever: Any | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 15.4 (1.9) [1.9 to 45.4]
  Fever: >=38.0 to 38.4 deg C | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 7.7 (0.2) [0.2 to 36.0]
  Fever: >38.4 to 38.9 deg C | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Fever: >38.9 to 40.0 deg C | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 7.7 (0.2) [0.2 to 36.0]
  Fever: >40.0 deg C | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Fatigue: Any | 22.2 (2.8) [2.8 to 60.0] | 6.7 (0.2) [0.2 to 31.9] | 7.7 (0.2) [0.2 to 36.0]
  Fatigue: Mild | 11.1 (0.3) [0.3 to 48.2] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Fatigue: Moderate | 11.1 (0.3) [0.3 to 48.2] | 6.7 (0.2) [0.2 to 31.9] | 7.7 (0.2) [0.2 to 36.0]
  Fatigue: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Fatigue: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Headache: Any | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Headache: Mild | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Headache: Moderate | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Headache: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Headache: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Chills: Any | 11.1 (0.3) [0.3 to 48.2] | 0 (0.0) [0.0 to 21.8] | 7.7 (0.2) [0.2 to 36.0]
  Chills: Mild | 11.1 (0.3) [0.3 to 48.2] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Chills: Moderate | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 7.7 (0.2) [0.2 to 36.0]
  Chills: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Chills: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Vomiting: Any | 11.1 (0.3) [0.3 to 48.2] | 0 (0.0) [0.0 to 21.8] | 23.1 (5.0) [5.0 to 53.8]
  Vomiting: Mild | 11.1 (0.3) [0.3 to 48.2] | 0 (0.0) [0.0 to 21.8] | 7.7 (0.2) [0.2 to 36.0]
  Vomiting: Moderate | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 15.4 (1.9) [1.9 to 45.4]
  Vomiting: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Vomiting: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Diarrhea: Any | 0 (0.0) [0.0 to 33.6] | 20.0 (4.3) [4.3 to 48.1] | 7.7 (0.2) [0.2 to 36.0]
  Diarrhea: Mild | 0 (0.0) [0.0 to 33.6] | 20.0 (4.3) [4.3 to 48.1] | 0 (0.0) [0.0 to 24.7]
  Diarrhea: Moderate | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  Diarrhea: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 7.7 (0.2) [0.2 to 36.0]
  Diarrhea: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  New or worsened muscle pain: Any | 11.1 (0.3) [0.3 to 48.2] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  New or worsened muscle pain: Mild | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  New or worsened muscle pain: Moderate | 11.1 (0.3) [0.3 to 48.2] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  New or worsened muscle pain: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  New or worsened muscle pain: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  New or worsened joint pain: Any | 11.1 (0.3) [0.3 to 48.2] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  New or worsened joint pain: Mild | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  New or worsened joint pain: Moderate | 11.1 (0.3) [0.3 to 48.2] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  New or worsened joint pain: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]
  New or worsened joint pain: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 24.7]

26. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 1 in Participants Aged >=5 to <12 Years
Description: Systemic events were recorded in an e-diary and at unscheduled clinical assessments from Day 1 to 7 after vaccination 1. Fever was defined as oral temperature >=38.0 deg C; categorised as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain: mild (did not interfere with activity), moderate (some interference with activity), severe (prevented daily routine activity).Vomiting: mild: 1-2 times in 24 hours, moderate: >2 times in 24 hours, severe: required intravenous hydration. Diarrhea: mild: 2-3 loose stools in 24 hours, moderate: 4-5 loose stools in 24 hours, severe: 6 or more loose stools in 24 hours. Grade 4 for all events: ER visit/hospitalization and were classified by investigator or medically qualified person. Events reported as AEs in the CRF within 7 days after vaccination were also included. Exact 95% CI based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 1
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 19 | 24 | 22
Percentage of participants
  Fever: Any | 0 [0.0 to 17.6] | 4.2 [0.1 to 21.1] | 0 [0.0 to 15.4]
  Fever: >=38.0 to 38.4 deg C | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Fever: >38.4 to 38.9 deg C | 0 [0.0 to 17.6] | 4.2 [0.1 to 21.1] | 0 [0.0 to 15.4]
  Fever: >38.9 to 40.0 deg C | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Fever: >40.0 deg C | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Fatigue: Any | 47.4 [24.4 to 71.1] | 37.5 [18.8 to 59.4] | 22.7 [7.8 to 45.4]
  Fatigue: Mild | 31.6 [12.6 to 56.6] | 20.8 [7.1 to 42.2] | 13.6 [2.9 to 34.9]
  Fatigue: Moderate | 15.8 [3.4 to 39.6] | 16.7 [4.7 to 37.4] | 9.1 [1.1 to 29.2]
  Fatigue: Severe | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Fatigue: Grade 4 | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Headache: Any | 42.1 [20.3 to 66.5] | 12.5 [2.7 to 32.4] | 22.7 [7.8 to 45.4]
  Headache: Mild | 31.6 [12.6 to 56.6] | 12.5 [2.7 to 32.4] | 9.1 [1.1 to 29.2]
  Headache: Moderate | 10.5 [1.3 to 33.1] | 0 [0.0 to 14.2] | 13.6 [2.9 to 34.9]
  Headache: Severe | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Headache: Grade 4 | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Chills: Any | 5.3 [0.1 to 26.0] | 0 [0.0 to 14.2] | 4.5 [0.1 to 22.8]
  Chills: Mild | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 4.5 [0.1 to 22.8]
  Chills: Moderate | 5.3 [0.1 to 26.0] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Chills: Severe | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Chills: Grade 4 | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Vomiting: Any | 5.3 [0.1 to 26.0] | 4.2 [0.1 to 21.1] | 0 [0.0 to 15.4]
  Vomiting: Mild | 5.3 [0.1 to 26.0] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Vomiting: Moderate | 0 [0.0 to 17.6] | 4.2 [0.1 to 21.1] | 0 [0.0 to 15.4]
  Vomiting: Severe | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Vomiting: Grade 4 | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Diarrhea: Any | 10.5 [1.3 to 33.1] | 0 [0.0 to 14.2] | 4.5 [0.1 to 22.8]
  Diarrhea: Mild | 10.5 [1.3 to 33.1] | 0 [0.0 to 14.2] | 4.5 [0.1 to 22.8]
  Diarrhea: Moderate | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Diarrhea: Severe | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  Diarrhea: Grade 4 | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  New or worsened muscle pain: Any | 5.3 [0.1 to 26.0] | 4.2 [0.1 to 21.1] | 0 [0.0 to 15.4]
  New or worsened muscle pain: Mild | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  New or worsened muscle pain: Moderate | 5.3 [0.1 to 26.0] | 4.2 [0.1 to 21.1] | 0 [0.0 to 15.4]
  New or worsened muscle pain: Severe | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  New or worsened joint pain: Any | 10.5 [1.3 to 33.1] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  New or worsened joint pain: Mild | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  New or worsened joint pain: Moderate | 10.5 [1.3 to 33.1] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  New or worsened joint pain: Severe | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 17.6] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4]

27. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 1 in Participants Aged >=12 to <18 Years
Description: as for outcome 26
Time Frame: Day 1 to Day 7 after Vaccination 1
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 7 | 1 | 7
Percentage of participants
  Fever: Any | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Fever: >=38.0 deg C to 38.4 deg C | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Fever: >38.4 deg C to 38.9 deg C | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Fever: >38.9 deg C to 40.0 deg C | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Fever: >40.0 deg C | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Fatigue: Any | 57.1 (18.4) [18.4 to 90.1] | 0 (0.0) [0.0 to 97.5] | 42.9 (9.9) [9.9 to 81.6]
  Fatigue: Mild | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 14.3 (0.4) [0.4 to 57.9]
  Fatigue: Moderate | 57.1 (18.4) [18.4 to 90.1] | 0 (0.0) [0.0 to 97.5] | 28.6 (3.7) [3.7 to 71.0]
  Fatigue: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Fatigue: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Headache: Any | 42.9 (9.9) [9.9 to 81.6] | 0 (0.0) [0.0 to 97.5] | 28.6 (3.7) [3.7 to 71.0]
  Headache: Mild | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 14.3 (0.4) [0.4 to 57.9]
  Headache: Moderate | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 97.5] | 14.3 (0.4) [0.4 to 57.9]
  Headache: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Headache: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Chills: Any | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Chills: Mild | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Chills: Moderate | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Chills: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Chills: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Vomiting: Any | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Vomiting: Mild | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Vomiting: Moderate | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Vomiting: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Vomiting: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Diarrhea: Any | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 28.6 (3.7) [3.7 to 71.0]
  Diarrhea: Mild | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 28.6 (3.7) [3.7 to 71.0]
  Diarrhea: Moderate | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Diarrhea: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  Diarrhea: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  New or worsened muscle pain: Any | 42.9 (9.9) [9.9 to 81.6] | 0 (0.0) [0.0 to 97.5] | 42.9 (9.9) [9.9 to 81.6]
  New or worsened muscle pain: Mild | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 42.9 (9.9) [9.9 to 81.6]
  New or worsened muscle pain: Moderate | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  New or worsened muscle pain: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  New or worsened muscle pain: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  New or worsened joint pain: Any | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  New or worsened joint pain: Mild | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  New or worsened joint pain: Moderate | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  New or worsened joint pain: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]
  New or worsened joint pain: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]

28. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 1 in Participants Aged >=18 Years
Description: as for outcome 26
Time Frame: Day 1 to Day 7 after Vaccination 1
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 5 | 1 | 1
Percentage of participants
  Fever: Any | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Fever: >=38.0 to 38.4 deg C | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Fever: >38.4 to 38.9 deg C | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Fever: >38.9 to 40.0 deg C | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Fever: >40.0 deg C | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Fatigue: Any | 60.0 [14.7 to 94.7] | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0]
  Fatigue: Mild | 40.0 [5.3 to 85.3] | 100.0 [2.5 to 100.0] | 0 [0.0 to 97.5]
  Fatigue: Moderate | 20.0 [0.5 to 71.6] | 0 [0.0 to 97.5] | 100.0 [2.5 to 100.0]
  Fatigue: Severe | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Fatigue: Grade 4 | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Headache: Any | 40.0 [5.3 to 85.3] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Headache: Mild | 20.0 [0.5 to 71.6] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Headache: Moderate | 20.0 [0.5 to 71.6] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Headache: Severe | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Headache: Grade 4 | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Chills: Any | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 100.0 [2.5 to 100.0]
  Chills: Mild | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 100.0 [2.5 to 100.0]
  Chills: Moderate | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Chills: Severe | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Chills: Grade 4 | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Vomiting: Any | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Vomiting: Mild | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Vomiting: Moderate | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Vomiting: Severe | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Vomiting: Grade 4 | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Diarrhea: Any | 40.0 [5.3 to 85.3] | 100.0 [2.5 to 100.0] | 0 [0.0 to 97.5]
  Diarrhea: Mild | 40.0 [5.3 to 85.3] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Diarrhea: Moderate | 0 [0.0 to 52.2] | 100.0 [2.5 to 100.0] | 0 [0.0 to 97.5]
  Diarrhea: Severe | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  Diarrhea: Grade 4 | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  New or worsened muscle pain: Any | 20.0 [0.5 to 71.6] | 100.0 [2.5 to 100.0] | 0 [0.0 to 97.5]
  New or worsened muscle pain: Mild | 0 [0.0 to 52.2] | 100.0 [2.5 to 100.0] | 0 [0.0 to 97.5]
  New or worsened muscle pain: Moderate | 20.0 [0.5 to 71.6] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  New or worsened muscle pain: Severe | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  New or worsened joint pain: Any | 20.0 [0.5 to 71.6] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  New or worsened joint pain: Mild | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  New or worsened joint pain: Moderate | 20.0 [0.5 to 71.6] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  New or worsened joint pain: Severe | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 52.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]

29. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 2 in Participants Aged >=2 to <5 Years
Description: Systemic events were recorded in an e-diary and at unscheduled clinical assessments from Day 1 to 7 after vaccination 2. Fever was defined as oral temperature >=38.0 deg C; categorised as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain: mild (did not interfere with activity), moderate (some interference with activity), severe (prevented daily routine activity).Vomiting: mild: 1-2 times in 24 hours, moderate: >2 times in 24 hours, severe: required intravenous hydration. Diarrhea: mild: 2-3 loose stools in 24 hours, moderate: 4-5 loose stools in 24 hours, severe: 6 or more loose stools in 24 hours. Grade 4 for all events: ER visit/hospitalization and were classified by investigator or medically qualified person. Events reported as AEs in the CRF within 7 days after vaccination were also included. Exact 95% CI based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 2
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 9 | 15 | 10
Percentage of participants
  Fever: Any | 11.1 [0.3 to 48.2] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Fever: >=38.0 deg C to 38.4 deg C | 11.1 [0.3 to 48.2] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Fever: >38.4 deg C to 38.9 deg C | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Fever: >38.9 deg C to 40.0 deg C | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Fever: >40.0 deg C | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Fatigue: Any | 0 [0.0 to 33.6] | 6.7 [0.2 to 31.9] | 10.0 [0.3 to 44.5]
  Fatigue: Mild | 0 [0.0 to 33.6] | 6.7 [0.2 to 31.9] | 10.0 [0.3 to 44.5]
  Fatigue: Moderate | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Fatigue: Severe | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Fatigue: Grade 4 | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Headache: Any | 0 [0.0 to 33.6] | 6.7 [0.2 to 31.9] | 0 [0.0 to 30.8]
  Headache: Mild | 0 [0.0 to 33.6] | 6.7 [0.2 to 31.9] | 0 [0.0 to 30.8]
  Headache: Moderate | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Headache: Severe | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Headache: Grade 4 | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Chills: Any | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Chills: Mild | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Chills: Moderate | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Chills: Severe | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Chills: Grade 4 | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Vomiting: Any | 0 [0.0 to 33.6] | 13.3 [1.7 to 40.5] | 10.0 [0.3 to 44.5]
  Vomiting: Mild | 0 [0.0 to 33.6] | 13.3 [1.7 to 40.5] | 0 [0.0 to 30.8]
  Vomiting: Moderate | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 10.0 [0.3 to 44.5]
  Vomiting: Severe | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Vomiting: Grade 4 | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Diarrhea: Any | 11.1 [0.3 to 48.2] | 6.7 [0.2 to 31.9] | 10.0 [0.3 to 44.5]
  Diarrhea: Mild | 11.1 [0.3 to 48.2] | 6.7 [0.2 to 31.9] | 10.0 [0.3 to 44.5]
  Diarrhea: Moderate | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Diarrhea: Severe | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  Diarrhea: Grade 4 | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  New or worsened muscle pain: Any | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  New or worsened muscle pain: Mild | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  New or worsened muscle pain: Moderate | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  New or worsened muscle pain: Severe | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  New or worsened joint pain: Any | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  New or worsened joint pain: Mild | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  New or worsened joint pain: Moderate | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  New or worsened joint pain: Severe | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 33.6] | 0 [0.0 to 21.8] | 0 [0.0 to 30.8]

30. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 2 in Participants Aged >=5 to <12 Years
Description: as for outcome 29
Time Frame: Day 1 to Day 7 after Vaccination 2
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 19 | 24 | 22
Percentage of participants
  Fever: Any | 5.3 (0.1) [0.1 to 26.0] | 0 (0.0) [0.0 to 14.2] | 4.5 (0.1) [0.1 to 22.8]
  Fever: >=38.0 deg C to 38.4 deg C | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Fever: >38.4 deg C to 38.9 deg C | 5.3 (0.1) [0.1 to 26.0] | 0 (0.0) [0.0 to 14.2] | 4.5 (0.1) [0.1 to 22.8]
  Fever: >38.9 deg C to 40.0 deg C | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Fever: >40.0 deg C | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Fatigue: Any | 57.9 (33.5) [33.5 to 79.7] | 37.5 (18.8) [18.8 to 59.4] | 45.5 (24.4) [24.4 to 67.8]
  Fatigue: Mild | 26.3 (9.1) [9.1 to 51.2] | 20.8 (7.1) [7.1 to 42.2] | 13.6 (2.9) [2.9 to 34.9]
  Fatigue: Moderate | 31.6 (12.6) [12.6 to 56.6] | 16.7 (4.7) [4.7 to 37.4] | 31.8 (13.9) [13.9 to 54.9]
  Fatigue: Severe | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Fatigue: Grade 4 | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Headache: Any | 36.8 (16.3) [16.3 to 61.6] | 29.2 (12.6) [12.6 to 51.1] | 18.2 (5.2) [5.2 to 40.3]
  Headache: Mild | 15.8 (3.4) [3.4 to 39.6] | 12.5 (2.7) [2.7 to 32.4] | 4.5 (0.1) [0.1 to 22.8]
  Headache: Moderate | 21.1 (6.1) [6.1 to 45.6] | 16.7 (4.7) [4.7 to 37.4] | 13.6 (2.9) [2.9 to 34.9]
  Headache: Severe | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Headache: Grade 4 | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Chills: Any | 21.1 (6.1) [6.1 to 45.6] | 4.2 (0.1) [0.1 to 21.1] | 4.5 (0.1) [0.1 to 22.8]
  Chills: Mild | 10.5 (1.3) [1.3 to 33.1] | 4.2 (0.1) [0.1 to 21.1] | 0 (0.0) [0.0 to 15.4]
  Chills: Moderate | 10.5 (1.3) [1.3 to 33.1] | 0 (0.0) [0.0 to 14.2] | 4.5 (0.1) [0.1 to 22.8]
  Chills: Severe | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Chills: Grade 4 | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Vomiting: Any | 0 (0.0) [0.0 to 17.6] | 12.5 (2.7) [2.7 to 32.4] | 0 (0.0) [0.0 to 15.4]
  Vomiting: Mild | 0 (0.0) [0.0 to 17.6] | 12.5 (2.7) [2.7 to 32.4] | 0 (0.0) [0.0 to 15.4]
  Vomiting: Moderate | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Vomiting: Severe | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Vomiting: Grade 4 | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Diarrhea: Any | 5.3 (0.1) [0.1 to 26.0] | 8.3 (1.0) [1.0 to 27.0] | 4.5 (0.1) [0.1 to 22.8]
  Diarrhea: Mild | 5.3 (0.1) [0.1 to 26.0] | 4.2 (0.1) [0.1 to 21.1] | 0 (0.0) [0.0 to 15.4]
  Diarrhea: Moderate | 0 (0.0) [0.0 to 17.6] | 4.2 (0.1) [0.1 to 21.1] | 4.5 (0.1) [0.1 to 22.8]
  Diarrhea: Severe | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  Diarrhea: Grade 4 | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  New or worsened muscle pain: Any | 10.5 (1.3) [1.3 to 33.1] | 12.5 (2.7) [2.7 to 32.4] | 4.5 (0.1) [0.1 to 22.8]
  New or worsened muscle pain: Mild | 0 (0.0) [0.0 to 17.6] | 4.2 (0.1) [0.1 to 21.1] | 0 (0.0) [0.0 to 15.4]
  New or worsened muscle pain: Moderate | 10.5 (1.3) [1.3 to 33.1] | 8.3 (1.0) [1.0 to 27.0] | 4.5 (0.1) [0.1 to 22.8]
  New or worsened muscle pain: Severe | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  New or worsened muscle pain: Grade 4 | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  New or worsened joint pain: Any | 15.8 (3.4) [3.4 to 39.6] | 4.2 (0.1) [0.1 to 21.1] | 4.5 (0.1) [0.1 to 22.8]
  New or worsened joint pain: Mild | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  New or worsened joint pain: Moderate | 15.8 (3.4) [3.4 to 39.6] | 4.2 (0.1) [0.1 to 21.1] | 4.5 (0.1) [0.1 to 22.8]
  New or worsened joint pain: Severe | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]
  New or worsened joint pain: Grade 4 | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 14.2] | 0 (0.0) [0.0 to 15.4]

31. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 2 in Participants Aged >=12 to <18 Years
Description: as for outcome 29
Time Frame: Day 1 to Day 7 after Vaccination 2
Population: Safety population consisted of all participants who received at least 1 dose of study intervention. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 7 | 1 | 6
Percentage of participants
  Fever: Any | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Fever: >=38.0 deg C to 38.4 deg C | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Fever: >38.4 deg C to 38.9 deg C | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Fever: >38.9 deg C to 40.0 deg C | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Fever: >40.0 deg C | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Fatigue: Any | 85.7 (42.1) [42.1 to 99.6] | 0 (0.0) [0.0 to 97.5] | 33.3 (4.3) [4.3 to 77.7]
  Fatigue: Mild | 42.9 (9.9) [9.9 to 81.6] | 0 (0.0) [0.0 to 97.5] | 33.3 (4.3) [4.3 to 77.7]
  Fatigue: Moderate | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Fatigue: Severe | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Fatigue: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Headache: Any | 71.4 (29.0) [29.0 to 96.3] | 0 (0.0) [0.0 to 97.5] | 16.7 (0.4) [0.4 to 64.1]
  Headache: Mild | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 97.5] | 16.7 (0.4) [0.4 to 64.1]
  Headache: Moderate | 42.9 (9.9) [9.9 to 81.6] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Headache: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Headache: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Chills: Any | 42.9 (9.9) [9.9 to 81.6] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Chills: Mild | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Chills: Moderate | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Chills: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Chills: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Vomiting: Any | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Vomiting: Mild | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Vomiting: Moderate | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Vomiting: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Vomiting: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Diarrhea: Any | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Diarrhea: Mild | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Diarrhea: Moderate | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Diarrhea: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  Diarrhea: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  New or worsened muscle pain: Any | 42.9 (9.9) [9.9 to 81.6] | 100.0 (2.5) [2.5 to 100.0] | 16.7 (0.4) [0.4 to 64.1]
  New or worsened muscle pain: Mild | 0 (0.0) [0.0 to 41.0] | 100.0 (2.5) [2.5 to 100.0] | 0 (0.0) [0.0 to 45.9]
  New or worsened muscle pain: Moderate | 42.9 (9.9) [9.9 to 81.6] | 0 (0.0) [0.0 to 97.5] | 16.7 (0.4) [0.4 to 64.1]
  New or worsened muscle pain: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  New or worsened muscle pain: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  New or worsened joint pain: Any | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  New or worsened joint pain: Mild | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  New or worsened joint pain: Moderate | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  New or worsened joint pain: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]
  New or worsened joint pain: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 45.9]

32. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 2 in Participants Aged >=18 Years
Description: as for outcome 29
Time Frame: Day 1 to Day 7 after Vaccination 2
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 5 | 1 | 1
Percentage of participants
  Fever: Any | 20.0 (0.5) [0.5 to 71.6] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Fever: >=38.0 to 38.4 deg C | 20.0 (0.5) [0.5 to 71.6] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Fever: >38.4 to 38.9 deg C | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Fever: >38.9 to 40.0 deg C | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Fever: >40.0 deg C | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Fatigue: Any | 60.0 (14.7) [14.7 to 94.7] | 100.0 (2.5) [2.5 to 100.0] | 0 (0.0) [0.0 to 97.5]
  Fatigue: Mild | 0 (0.0) [0.0 to 52.2] | 100.0 (2.5) [2.5 to 100.0] | 0 (0.0) [0.0 to 97.5]
  Fatigue: Moderate | 60.0 (14.7) [14.7 to 94.7] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Fatigue: Severe | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Fatigue: Grade 4 | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Headache: Any | 60.0 (14.7) [14.7 to 94.7] | 100.0 (2.5) [2.5 to 100.0] | 0 (0.0) [0.0 to 97.5]
  Headache: Mild | 20.0 (0.5) [0.5 to 71.6] | 100.0 (2.5) [2.5 to 100.0] | 0 (0.0) [0.0 to 97.5]
  Headache: Moderate | 40.0 (5.3) [5.3 to 85.3] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Headache: Severe | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Headache: Grade 4 | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Chills: Any | 40.0 (5.3) [5.3 to 85.3] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Chills: Mild | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Chills: Moderate | 40.0 (5.3) [5.3 to 85.3] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Chills: Severe | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Chills: Grade 4 | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Vomiting: Any | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Vomiting: Mild | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Vomiting: Moderate | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Vomiting: Severe | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Vomiting: Grade 4 | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Diarrhea: Any | 60.0 (14.7) [14.7 to 94.7] | 100.0 (2.5) [2.5 to 100.0] | 0 (0.0) [0.0 to 97.5]
  Diarrhea: Mild | 40.0 (5.3) [5.3 to 85.3] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Diarrhea: Moderate | 20.0 (0.5) [0.5 to 71.6] | 100.0 (2.5) [2.5 to 100.0] | 0 (0.0) [0.0 to 97.5]
  Diarrhea: Severe | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  Diarrhea: Grade 4 | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  New or worsened muscle pain: Any | 20.0 (0.5) [0.5 to 71.6] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  New or worsened muscle pain: Mild | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  New or worsened muscle pain: Moderate | 20.0 (0.5) [0.5 to 71.6] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  New or worsened muscle pain: Severe | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  New or worsened muscle pain: Grade 4 | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  New or worsened joint pain: Any | 20.0 (0.5) [0.5 to 71.6] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  New or worsened joint pain: Mild | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  New or worsened joint pain: Moderate | 20.0 (0.5) [0.5 to 71.6] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  New or worsened joint pain: Severe | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]
  New or worsened joint pain: Grade 4 | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]

33. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 3 in Participants Aged >=2 to <5 Years
Description: Systemic events were recorded in an e-diary and at unscheduled clinical assessments from Day 1 to 7 after vaccination 3. Fever was defined as oral temperature >=38.0 deg C; categorised as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain: mild (did not interfere with activity), moderate (some interference with activity), severe (prevented daily routine activity).Vomiting: mild: 1-2 times in 24 hours, moderate: >2 times in 24 hours, severe: required intravenous hydration. Diarrhea: mild: 2-3 loose stools in 24 hours, moderate: 4-5 loose stools in 24 hours, severe: 6 or more loose stools in 24 hours. Grade 4 for all events: ER visit/hospitalization and were classified by investigator or medically qualified person. Events reported as AEs in the CRF within 7 days after vaccination were also included. Exact 95% CI based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 3
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 9 | 15 | 11
Percentage of participants
  Fever: Any | 0 (0.0) [0.0 to 33.6] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 28.5]
  Fever: >=38.0 deg C to 38.4 deg C | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Fever: >38.4 deg C to 38.9 deg C | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Fever: >38.9 deg C to 40.0 deg C | 0 (0.0) [0.0 to 33.6] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 28.5]
  Fever: >40.0 deg C | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Fatigue: Any | 11.1 (0.3) [0.3 to 48.2] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 28.5]
  Fatigue: Mild | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Fatigue: Moderate | 11.1 (0.3) [0.3 to 48.2] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 28.5]
  Fatigue: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Fatigue: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Headache: Any | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Headache: Mild | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Headache: Moderate | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Headache: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Headache: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Chills: Any | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Chills: Mild | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Chills: Moderate | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Chills: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Chills: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Vomiting: Any | 0 (0.0) [0.0 to 33.6] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 28.5]
  Vomiting: Mild | 0 (0.0) [0.0 to 33.6] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 28.5]
  Vomiting: Moderate | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Vomiting: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Vomiting: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Diarrhea: Any | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Diarrhea: Mild | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Diarrhea: Moderate | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Diarrhea: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  Diarrhea: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  New or worsened muscle pain: Any | 0 (0.0) [0.0 to 33.6] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 28.5]
  New or worsened muscle pain: Mild | 0 (0.0) [0.0 to 33.6] | 6.7 (0.2) [0.2 to 31.9] | 0 (0.0) [0.0 to 28.5]
  New or worsened muscle pain: Moderate | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  New or worsened muscle pain: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  New or worsened muscle pain: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  New or worsened joint pain: Any | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  New or worsened joint pain: Mild | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  New or worsened joint pain: Moderate | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  New or worsened joint pain: Severe | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]
  New or worsened joint pain: Grade 4 | 0 (0.0) [0.0 to 33.6] | 0 (0.0) [0.0 to 21.8] | 0 (0.0) [0.0 to 28.5]

34. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 3 in Participants Aged >=5 to <12 Years
Description: as for outcome 33
Time Frame: Day 1 to Day 7 after Vaccination 3
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 17 | 23 | 21
Percentage of participants
  Fever: Any | 17.6 [3.8 to 43.4] | 0 [0.0 to 14.8] | 19.0 [5.4 to 41.9]
  Fever: >=38.0 to 38.4 deg C | 11.8 [1.5 to 36.4] | 0 [0.0 to 14.8] | 14.3 [3.0 to 36.3]
  Fever: >38.4 to 38.9 deg C | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  Fever: >38.9 to 40.0 deg C | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 4.8 [0.1 to 23.8]
  Fever: >40.0 deg C | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  Fever: Unknown | 5.9 [0.1 to 28.7] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  Fatigue: Any | 47.1 [23.0 to 72.2] | 34.8 [16.4 to 57.3] | 52.4 [29.8 to 74.3]
  Fatigue: Mild | 35.3 [14.2 to 61.7] | 13.0 [2.8 to 33.6] | 23.8 [8.2 to 47.2]
  Fatigue: Moderate | 11.8 [1.5 to 36.4] | 21.7 [7.5 to 43.7] | 28.6 [11.3 to 52.2]
  Fatigue: Severe | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  Fatigue: Grade 4 | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  Headache: Any | 35.3 [14.2 to 61.7] | 8.7 [1.1 to 28.0] | 28.6 [11.3 to 52.2]
  Headache: Mild | 29.4 [10.3 to 56.0] | 4.3 [0.1 to 21.9] | 9.5 [1.2 to 30.4]
  Headache: Moderate | 5.9 [0.1 to 28.7] | 0 [0.0 to 14.8] | 19.0 [5.4 to 41.9]
  Headache: Severe | 0 [0.0 to 19.5] | 4.3 [0.1 to 21.9] | 0 [0.0 to 16.1]
  Headache: Grade 4 | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  Chills: Any | 17.6 [3.8 to 43.4] | 4.3 [0.1 to 21.9] | 14.3 [3.0 to 36.3]
  Chills: Mild | 5.9 [0.1 to 28.7] | 4.3 [0.1 to 21.9] | 4.8 [0.1 to 23.8]
  Chills: Moderate | 11.8 [1.5 to 36.4] | 0 [0.0 to 14.8] | 9.5 [3.0 to 36.3]
  Chills: Severe | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  Chills: Grade 4 | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  Vomiting: Any | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 4.8 [0.1 to 23.8]
  Vomiting: Mild | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  Vomiting: Moderate | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 4.8 [0.1 to 23.8]
  Vomiting: Severe | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  Vomiting: Grade 4 | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  Diarrhea: Any | 11.8 [1.5 to 36.4] | 0 [0.0 to 14.8] | 4.8 [0.1 to 23.8]
  Diarrhea: Mild | 11.8 [1.5 to 36.4] | 0 [0.0 to 14.8] | 4.8 [0.1 to 23.8]
  Diarrhea: Moderate | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  Diarrhea: Severe | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  Diarrhea: Grade 4 | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  New or worsened muscle pain: Any | 29.4 [10.3 to 56.0] | 13.0 [2.8 to 33.6] | 4.8 [0.1 to 23.8]
  New or worsened muscle pain: Mild | 5.9 [0.1 to 28.7] | 13.0 [2.8 to 33.6] | 4.8 [0.1 to 23.8]
  New or worsened muscle pain: Moderate | 23.5 [6.8 to 49.9] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  New or worsened muscle pain: Severe | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  New or worsened joint pain: Any | 11.8 [1.5 to 36.4] | 4.3 [2.8 to 33.6] | 4.8 [0.1 to 23.8]
  New or worsened joint pain: Mild | 0 [0.0 to 19.5] | 4.3 [2.8 to 33.6] | 4.8 [0.1 to 23.8]
  New or worsened joint pain: Moderate | 11.8 [1.5 to 36.4] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  New or worsened joint pain: Severe | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 19.5] | 0 [0.0 to 14.8] | 0 [0.0 to 16.1]

35. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 3 in Participants Aged >=12 to <18 Years
Description: as for outcome 33
Time Frame: Day 1 to Day 7 after Vaccination 3
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 7 | 1 | 6
Percentage of participants
  Fever: Any | 42.9 [9.9 to 81.6] | 0 [0.0 to 97.5] | 33.3 [4.3 to 77.7]
  Fever: >=38.0 to 38.4 deg C | 28.6 [3.7 to 71.0] | 0 [0.0 to 97.5] | 33.3 [4.3 to 77.7]
  Fever: >38.4°C to 38.9 deg C | 14.3 [0.4 to 57.9] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Fever: >38.9°C to 40.0 deg C | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Fever: >40.0 deg C | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Fatigue: Any | 85.7 [42.1 to 99.6] | 100.0 [2.5 to 100.0] | 50.0 [11.8 to 88.2]
  Fatigue: Mild | 14.3 [0.4 to 57.9] | 100.0 [2.5 to 100.0] | 50.0 [11.8 to 88.2]
  Fatigue: Moderate | 71.4 [29.0 to 96.3] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Fatigue: Severe | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Fatigue: Grade 4 | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Headache: Any | 85.7 [42.1 to 99.6] | 100.0 [2.5 to 100.0] | 66.7 [22.3 to 95.7]
  Headache: Mild | 28.6 [3.7 to 71.0] | 100.0 [2.5 to 100.0] | 33.3 [4.3 to 77.7]
  Headache: Moderate | 57.1 [18.4 to 90.1] | 0 [0.0 to 97.5] | 33.3 [4.3 to 77.7]
  Headache: Severe | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Headache: Grade 4 | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Chills: Any | 71.4 [29.0 to 96.3] | 100.0 [2.5 to 100.0] | 16.7 [0.4 to 64.1]
  Chills: Mild | 14.3 [0.4 to 57.9] | 100.0 [2.5 to 100.0] | 16.7 [0.4 to 64.1]
  Chills: Moderate | 57.1 [18.4 to 90.1] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Chills: Severe | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Chills: Grade 4 | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Vomiting: Any | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Vomiting: Mild | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Vomiting: Moderate | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Vomiting: Severe | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Vomiting: Grade 4 | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Diarrhea: Any | 14.3 [0.4 to 57.9] | 0 [0.0 to 97.5] | 33.3 [4.3 to 77.7]
  Diarrhea: Mild | 14.3 [0.4 to 57.9] | 0 [0.0 to 97.5] | 33.3 [4.3 to 77.7]
  Diarrhea: Moderate | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Diarrhea: Severe | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  Diarrhea: Grade 4 | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  New or worsened muscle pain: Any | 28.6 [3.7 to 71.0] | 0 [0.0 to 97.5] | 16.7 [0.4 to 64.1]
  New or worsened muscle pain: Mild | 14.3 [0.4 to 57.9] | 0 [0.0 to 97.5] | 16.7 [0.4 to 64.1]
  New or worsened muscle pain: Moderate | 14.3 [0.4 to 57.9] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  New or worsened muscle pain: Severe | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  New or worsened joint pain: Any | 14.3 [0.4 to 57.9] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  New or worsened joint pain: Mild | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  New or worsened joint pain: Moderate | 14.3 [0.4 to 57.9] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  New or worsened joint pain: Severe | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 41.0] | 0 [0.0 to 97.5] | 0 [0.0 to 45.9]

36. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 3 in Participants Aged >=18 Years
Description: as for outcome 33
Time Frame: Day 1 to Day 7 after Vaccination 3
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 4 | 0 | 1
Percentage of participants
  Fever:Any | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Fever: >=38.0 to 38.4 deg C | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Fever: >38.4 to 38.9 deg C | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Fever: >38.9 to 40.0 deg C | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Fever: >40.0 deg C | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Fatigue: Any | 75.0 [19.4 to 99.4] |  | 0 [0.0 to 97.5]
  Fatigue: Mild | 50.0 [6.8 to 93.2] |  | 0 [0.0 to 97.5]
  Fatigue: Moderate | 25.0 [0.6 to 80.6] |  | 0 [0.0 to 97.5]
  Fatigue: Severe | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Fatigue: Grade 4 | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Headache: Any | 75.0 [19.4 to 99.4] |  | 0 [0.0 to 97.5]
  Headache: Mild | 25.0 [0.6 to 80.6] |  | 0 [0.0 to 97.5]
  Headache: Moderate | 50.0 [6.8 to 93.2] |  | 0 [0.0 to 97.5]
  Headache: Severe | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Headache: Grade 4 | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Chills: Any | 50.0 [6.8 to 93.2] |  | 0 [0.0 to 97.5]
  Chills: Mild | 25.0 [0.6 to 80.6] |  | 0 [0.0 to 97.5]
  Chills: Moderate | 25.0 [0.6 to 80.6] |  | 0 [0.0 to 97.5]
  Chills: Severe | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Chills: Grade 4 | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Vomiting: Any | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Vomiting: Mild | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Vomiting: Moderate | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Vomiting: Severe | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Vomiting: Grade 4 | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Diarrhea: Any | 25.0 [0.6 to 80.6] |  | 0 [0.0 to 97.5]
  Diarrhea: Mild | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Diarrhea: Moderate | 25.0 [0.6 to 80.6] |  | 0 [0.0 to 97.5]
  Diarrhea: Severe | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  Diarrhea: Grade 4 | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  New or worsened muscle pain: Any | 50.0 [6.8 to 93.2] |  | 0 [0.0 to 97.5]
  New or worsened muscle pain: Mild | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  New or worsened muscle pain: Moderate | 50.0 [6.8 to 93.2] |  | 0 [0.0 to 97.5]
  New or worsened muscle pain: Severe | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  New or worsened joint pain: Any | 50.0 [6.8 to 93.2] |  | 0 [0.0 to 97.5]
  New or worsened joint pain: Mild | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  New or worsened joint pain: Moderate | 50.0 [6.8 to 93.2] |  | 0 [0.0 to 97.5]
  New or worsened joint pain: Severe | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 60.2] |  | 0 [0.0 to 97.5]

37. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 4 in Participants Aged >=2 to <5 Years
Description: Systemic events were recorded in an e-diary and at unscheduled clinical assessments from Day 1 to 7 after vaccination 4. Fever was defined as oral temperature >=38.0 deg C; categorised as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain: mild (did not interfere with activity), moderate (some interference with activity), severe (prevented daily routine activity).Vomiting: mild: 1-2 times in 24 hours, moderate: >2 times in 24 hours, severe: required intravenous hydration. Diarrhea: mild: 2-3 loose stools in 24 hours, moderate: 4-5 loose stools in 24 hours, severe: 6 or more loose stools in 24 hours. Grade 4 for all events: ER visit/hospitalization and were classified by investigator or medically qualified person. Events reported as AEs in the CRF within 7 days after vaccination were also included. Exact 95% CI based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 4
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 7 | 6 | 6
Percentage of participants
  Fever: Any | 28.6 (3.7) [3.7 to 71.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Fever: >=38.0 to 38.4 deg C | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Fever: >38.4 to 38.9 deg C | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Fever: >38.9 to 40.0 deg C | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Fever: >40.0 deg C | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Fatigue: Any | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 45.9] | 16.7 (0.4) [0.4 to 64.1]
  Fatigue: Mild | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 45.9] | 16.7 (0.4) [0.4 to 64.1]
  Fatigue: Moderate | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Fatigue: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Fatigue: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Headache: Any | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Headache: Mild | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Headache: Moderate | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Headache: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Headache: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Chills: Any | 14.3 (0.4) [0.4 to 57.9] | 16.7 (0.4) [0.4 to 64.1] | 0 (0.0) [0.0 to 45.9]
  Chills: Mild | 0 (0.0) [0.0 to 41.0] | 16.7 (0.4) [0.4 to 64.1] | 0 (0.0) [0.0 to 45.9]
  Chills: Moderate | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Chills: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Chills: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Vomiting: Any | 0 (0.0) [0.0 to 41.0] | 16.7 (0.4) [0.4 to 64.1] | 0 (0.0) [0.0 to 45.9]
  Vomiting: Mild | 0 (0.0) [0.0 to 41.0] | 16.7 (0.4) [0.4 to 64.1] | 0 (0.0) [0.0 to 45.9]
  Vomiting: Moderate | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Vomiting: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Vomiting: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Diarrhea: Any | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Diarrhea: Mild | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Diarrhea: Moderate | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Diarrhea: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  Diarrhea: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  New or worsened muscle pain: Any | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  New or worsened muscle pain: Mild | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  New or worsened muscle pain: Moderate | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  New or worsened muscle pain: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  New or worsened muscle pain: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  New or worsened joint pain: Any | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  New or worsened joint pain: Mild | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  New or worsened joint pain: Moderate | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  New or worsened joint pain: Severe | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]
  New or worsened joint pain: Grade 4 | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 45.9] | 0 (0.0) [0.0 to 45.9]

38. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 4 in Participants Aged >=5 to <12 Years
Description: Systemic events were recorded in an e-diary and at unscheduled clinical assessments from Day 1 to 7 after vaccination 4. Fever was defined as oral temperature >=38.0 deg C; categorised as >=38.0 to 38.4 deg C, >38.4 to 38.9 de, >38.9 to 40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain: mild (did not interfere with activity), moderate (some interference with activity), severe (prevented daily routine activity).Vomiting: mild: 1-2 times in 24 hours, moderate: >2 times in 24 hours, severe: required intravenous hydration. Diarrhea: mild: 2-3 loose stools in 24 hours, moderate: 4-5 loose stools in 24 hours, severe: 6 or more loose stools in 24 hours. Grade 4 for all events: ER visit/hospitalization and were classified by investigator or medically qualified person. Events reported as AEs in the CRF within 7 days after vaccination were also included. Exact 95% CI based on Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after Vaccination 4
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 12 | 19 | 15
Percentage of participants
  Fever: Any | 8.3 (0.2) [0.2 to 38.5] | 5.3 (0.1) [0.1 to 26.0] | 6.7 (0.2) [0.2 to 31.9]
  Fever: >=38.0 to 38.4 deg C | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Fever: >38.4 to 38.9 deg C | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Fever: >38.9 to 40.0 deg C | 8.3 (0.2) [0.2 to 38.5] | 5.3 (0.1) [0.1 to 26.0] | 6.7 (0.2) [0.2 to 31.9]
  Fever: >40.0 deg C | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Fatigue: Any | 50.0 (21.1) [21.1 to 78.9] | 26.3 (9.1) [9.1 to 51.2] | 33.3 (11.8) [11.8 to 61.6]
  Fatigue: Mild | 33.3 (9.9) [9.9 to 65.1] | 10.5 (1.3) [1.3 to 33.1] | 13.3 (1.7) [1.7 to 40.5]
  Fatigue: Moderate | 16.7 (2.1) [2.1 to 48.4] | 15.8 (3.4) [3.4 to 39.6] | 20.0 (4.3) [4.3 to 48.1]
  Fatigue: Severe | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Fatigue: Grade 4 | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Headache: Any | 33.3 (9.9) [9.9 to 65.1] | 21.1 (6.1) [6.1 to 45.6] | 13.3 (1.7) [1.7 to 40.5]
  Headache: Mild | 8.3 (0.2) [0.2 to 38.5] | 15.8 (3.4) [3.4 to 39.6] | 0 (0.0) [0.0 to 21.8]
  Headache: Moderate | 25.0 (5.5) [5.5 to 57.2] | 5.3 (0.1) [0.1 to 26.0] | 6.7 (0.2) [0.2 to 31.9]
  Headache: Severe | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 6.7 (0.2) [0.2 to 31.9]
  Headache: Grade 4 | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Chills: Any | 8.3 (0.2) [0.2 to 38.5] | 5.3 (0.1) [0.1 to 26.0] | 13.3 (1.7) [1.7 to 40.5]
  Chills: Mild | 8.3 (0.2) [0.2 to 38.5] | 5.3 (0.1) [0.1 to 26.0] | 0 (0.0) [0.0 to 21.8]
  Chills: Moderate | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 13.3 (1.7) [1.7 to 40.5]
  Chills: Severe | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Chills: Grade 4 | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Vomiting: Any | 8.3 (0.2) [0.2 to 38.5] | 5.3 (0.1) [0.1 to 26.0] | 0 (0.0) [0.0 to 21.8]
  Vomiting: Mild | 8.3 (0.2) [0.2 to 38.5] | 5.3 (0.1) [0.1 to 26.0] | 0 (0.0) [0.0 to 21.8]
  Vomiting: Moderate | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Vomiting: Severe | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Vomiting: Grade 4 | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Diarrhea: Any | 25.0 (5.5) [5.5 to 57.2] | 15.8 (3.4) [3.4 to 39.6] | 6.7 (0.2) [0.2 to 31.9]
  Diarrhea: Mild | 25.0 (5.5) [5.5 to 57.2] | 10.5 (1.3) [1.3 to 33.1] | 6.7 (0.2) [0.2 to 31.9]
  Diarrhea: Moderate | 0 (0.0) [0.0 to 26.5] | 5.3 (0.1) [0.1 to 26.0] | 0 (0.0) [0.0 to 21.8]
  Diarrhea: Severe | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  Diarrhea: Grade 4 | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  New or worsened muscle pain: Any | 16.7 (2.1) [2.1 to 48.4] | 15.8 (3.4) [3.4 to 39.6] | 6.7 (0.2) [0.2 to 31.9]
  New or worsened muscle pain: Mild | 0 (0.0) [0.0 to 26.5] | 15.8 (3.4) [3.4 to 39.6] | 0 (0.0) [0.0 to 21.8]
  New or worsened muscle pain: Moderate | 8.3 (0.2) [0.2 to 38.5] | 0 (0.0) [0.0 to 17.6] | 6.7 (0.2) [0.2 to 31.9]
  New or worsened muscle pain: Severe | 8.3 (0.2) [0.2 to 38.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  New or worsened muscle pain: Grade 4 | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  New or worsened joint pain: Any | 25.0 (5.5) [5.5 to 57.2] | 0 (0.0) [0.0 to 17.6] | 6.7 (0.2) [0.2 to 31.9]
  New or worsened joint pain: Mild | 8.3 (0.2) [0.2 to 38.5] | 0 (0.0) [0.0 to 17.6] | 6.7 (0.2) [0.2 to 31.9]
  New or worsened joint pain: Moderate | 16.7 (2.1) [2.1 to 48.4] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  New or worsened joint pain: Severe | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]
  New or worsened joint pain: Grade 4 | 0 (0.0) [0.0 to 26.5] | 0 (0.0) [0.0 to 17.6] | 0 (0.0) [0.0 to 21.8]

39. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 4 in Participants Aged >=12 to <18 Years
Description: as for outcome 37
Time Frame: Day 1 to Day 7 after Vaccination 4
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 4 | 1 | 3
Percentage of participants
  Fever: Any | 25.0 [0.6 to 80.6] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Fever: >=38.0 to 38.4 deg C | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Fever: >38.4 to 38.9 deg C | 25.0 [0.6 to 80.6] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Fever: >38.9 to 40.0 deg C | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Fever: >40.0 deg C | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Fatigue: Any | 50.0 [6.8 to 93.2] | 100.0 [2.5 to 100.0] | 66.7 [9.4 to 99.2]
  Fatigue: Mild | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Fatigue: Moderate | 50.0 [6.8 to 93.2] | 100.0 [2.5 to 100.0] | 33.3 [0.8 to 90.6]
  Fatigue: Severe | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Fatigue: Grade 4 | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Headache: Any | 25.0 [0.6 to 80.6] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Headache: Mild | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Headache: Moderate | 25.0 [0.6 to 80.6] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Headache: Severe | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Headache: Grade 4 | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Chills: Any | 25.0 [0.6 to 80.6] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Chills: Mild | 25.0 [0.6 to 80.6] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Chills: Moderate | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Chills: Severe | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Chills: Grade 4 | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Vomiting: Any | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Vomiting: Mild | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Vomiting: Moderate | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Vomiting: Severe | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Vomiting: Grade 4 | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Diarrhea: Any | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Diarrhea: Mild | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Diarrhea: Moderate | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  Diarrhea: Severe | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  Diarrhea: Grade 4 | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  New or worsened muscle pain: Any | 25.0 [0.6 to 80.6] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  New or worsened muscle pain: Mild | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  New or worsened muscle pain: Moderate | 25.0 [0.6 to 80.6] | 0 [0.0 to 97.5] | 33.3 [0.8 to 90.6]
  New or worsened muscle pain: Severe | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5]
  New or worsened joint pain: Any | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  New or worsened joint pain: Mild | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  New or worsened joint pain: Moderate | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  New or worsened joint pain: Severe | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 60.2] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8]

40. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 4 in Participants Aged >=18 Years
Description: as for outcome 37
Time Frame: Day 1 to Day 7 after Vaccination 4
Population: Safety population consisted of all participants who received at least 1 dose of study intervention.Here, 'Overall Number of Participants Analyzed (N)' signifies participants evaluable for this outcome measure. Participants of >=18 years Haemodialysis: group did not receive Vaccination 4 and therefore were not analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 3 | 1 | 0
Percentage of participants
  Fever: Any | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Fever: >=38.0 to 38.4 deg C | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Fever: >38.4 to 38.9 deg C | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Fever: >38.9 to 40.0 deg C | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Fever: >40.0 deg C | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Fatigue: Any | 66.7 (9.4) [9.4 to 99.2] | 0 (0.0) [0.0 to 97.5] |
  Fatigue: Mild | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  Fatigue: Moderate | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  Fatigue: Severe | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Fatigue: Grade 4 | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Headache: Any | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  Headache: Mild | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  Headache: Moderate | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Headache: Severe | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Headache: Grade 4 | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Chills: Any | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  Chills: Mild | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Chills: Moderate | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  Chills: Severe | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Chills: Grade 4 | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Vomiting: Any | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Vomiting: Mild | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Vomiting: Moderate | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Vomiting: Severe | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Vomiting: Grade 4 | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Diarrhea: Any | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Diarrhea: Mild | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Diarrhea: Moderate | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Diarrhea: Severe | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  Diarrhea: Grade 4 | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  New or worsened muscle pain: Any | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  New or worsened muscle pain: Mild | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  New or worsened muscle pain: Moderate | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  New or worsened muscle pain: Severe | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  New or worsened muscle pain: Grade 4 | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  New or worsened joint pain: Any | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  New or worsened joint pain: Mild | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  New or worsened joint pain: Moderate | 33.3 (0.8) [0.8 to 90.6] | 0 (0.0) [0.0 to 97.5] |
  New or worsened joint pain: Severe | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |
  New or worsened joint pain: Grade 4 | 0 (0.0) [0.0 to 70.8] | 0 (0.0) [0.0 to 97.5] |

41. Primary Outcome: Percentage of Participants Reporting at Least 1 Adverse Event (AE) After Vaccination 1 to 1 Month After Vaccination 2 in Participants Aged >=2 to <5 Years
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants reporting AEs after vaccination 1 to 1 month after vaccination 2 were reported in this outcome measure. Exact 2-sided CI based on the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From Vaccination 1 to 1 month after Vaccination 2
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 9 | 15 | 13
Percentage of participants | 44.4 (13.7) [13.7 to 78.8] | 33.3 (11.8) [11.8 to 61.6] | 38.5 (13.9) [13.9 to 68.4]

42. Primary Outcome: Percentage of Participants Reporting at Least 1 Adverse Event After Vaccination 1 to 1 Month After Vaccination 2 in Participants Aged >=5 to <12 Years
Description: as for outcome 41
Time Frame: From Vaccination 1 to 1 month after Vaccination 2
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 19 | 24 | 22
Percentage of participants | 36.8 [16.3 to 61.6] | 8.3 [1.0 to 27.0] | 27.3 [10.7 to 50.2]

43. Primary Outcome: Percentage of Participants Reporting at Least 1 Adverse Event After Vaccination 1 to 1 Month After Vaccination 2 in Participants Aged >=12 to <18 Years
Description: as for outcome 41
Time Frame: From Vaccination 1 to 1 month after Vaccination 2
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 7 | 1 | 7
Percentage of participants | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 14.3 (0.4) [0.4 to 57.9]

44. Primary Outcome: Percentage of Participants Reporting at Least 1 Adverse Event After Vaccination 1 to 1 Month After Vaccination 2 in Participants Aged >=18 Years
Description: as for outcome 41
Time Frame: From Vaccination 1 to 1 month after Vaccination 2
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 5 | 1 | 1
Percentage of participants | 20.0 (0.5) [0.5 to 71.6] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]

45. Primary Outcome: Percentage of Participants Reporting at Least 1 Adverse Event From Vaccination 3 to 1 Month After Vaccination 3 in Participants Aged >=2 to <5 Years
Description: as for outcome 41
Time Frame: From Vaccination 3 to 1 month after Vaccination 3
Population: Safety population included all participants who received at least 1 dose of the study intervention. Here, Overall Number of Participants Analyzed signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 9 | 15 | 11
Percentage of participants | 33.3 (7.5) [7.5 to 70.1] | 40.0 (16.3) [16.3 to 67.7] | 0 (0.0) [0.0 to 28.5]

46. Primary Outcome: Percentage of Participants Reporting at Least 1 Adverse Event From Vaccination 3 to 1 Month After Vaccination 3 in Participants Aged >=5 to <12 Years
Description: as for outcome 41
Time Frame: From Vaccination 3 to 1 month after Vaccination 3
Population: as for outcome 45
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 17 | 23 | 22
Percentage of participants | 29.4 (10.3) [10.3 to 56.0] | 8.7 (1.1) [1.1 to 28.0] | 4.5 (0.1) [0.1 to 22.8]

47. Primary Outcome: Percentage of Participants Reporting at Least 1 Adverse Event From Vaccination 3 to 1 Month After Vaccination 3 in Participants Aged >=12 to <18 Years
Description: as for outcome 41
Time Frame: From Vaccination 3 to 1 month after Vaccination 3
Population: as for outcome 45
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 7 | 1 | 6
Percentage of participants | 14.3 (0.4) [0.4 to 57.9] | 0 (0.0) [0.0 to 97.5] | 16.7 (0.4) [0.4 to 64.1]

48. Primary Outcome: Percentage of Participants Reporting at Least 1 Adverse Event After Vaccination 3 to 1 Month After Vaccination 3 in Participants Aged >=18 Years
Description: as for outcome 41
Time Frame: From Vaccination 3 to 1 month after Vaccination 3
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 5 | 1 | 1
Percentage of participants | 0 (0.0) [0.0 to 52.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 97.5]

49. Primary Outcome: Percentage of Participants Reporting at Least 1 Adverse Event From Vaccination 4 to 1 Month After Vaccination 4 in Participants Aged >=2 to <5 Years
Description: as for outcome 41
Time Frame: From Vaccination 4 to 1 month after Vaccination 4
Population: Safety population included all participants who received at least 1 dose of the study intervention. Here, 'Overall Number of Participants Analyzed (N)' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 7 | 6 | 6
Percentage of participants | 14.3 (0.4) [0.4 to 57.9] | 16.7 (0.4) [0.4 to 64.1] | 0 (0.0) [0.0 to 45.9]

50. Primary Outcome: Percentage of Participants Reporting at Least 1 Adverse Event From Vaccination 4 to 1 Month After Vaccination 4 in Participants Aged >=5 to <12 Years
Description: as for outcome 41
Time Frame: From Vaccination 4 to 1 month after Vaccination 4
Population: as for outcome 49
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 12 | 19 | 15
Percentage of participants | 0 (0.0) [0.0 to 26.5] | 36.8 (16.3) [16.3 to 61.6] | 0 (0.0) [0.0 to 21.8]

51. Primary Outcome: Percentage of Participants Reporting at Least 1 Adverse Event From Vaccination 4 to 1 Month After Vaccination 4 in Participants Aged >=12 to <18 Years
Description: as for outcome 41
Time Frame: From Vaccination 4 to 1 month after Vaccination 4
Population: as for outcome 49
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 4 | 1 | 3
Percentage of participants | 0 (0.0) [0.0 to 60.2] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 70.8]

52. Primary Outcome: Percentage of Participants Reporting at Least 1 Adverse Event After Vaccination 4 to 1 Month After Vaccination 4 in Participants Aged >=18 Years
Description: as for outcome 41
Time Frame: From Vaccination 4 to 1 month after Vaccination 4
Population: Safety population included all participants who received at least 1 dose of the study intervention. Here, Overall Number of Participants Analyzed signifies participants evaluable for this outcome measure.Participants of >=18 years with Haemodialysis: group did not receive Vaccination 4 and therefore were not analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 3 | 1 | 0
Percentage of participants | 0 (0.0) [0.0 to 70.8] | 100.0 (2.5) [2.5 to 100.0] |

53. Primary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs) From Vaccination 1 Through the Duration of the Study in Participants Aged >=2 to <5 Years
Description: An SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening; resulted in persistent disability/incapacity; constituted a congenital anomaly/birth defect; was important medical event; required inpatient hospitalization or prolongation of existing hospitalization, was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic, and other situations as medical judgement of investigator. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: From Vaccination 1 to 6 months after Vaccination 4 (approximately 14 months)
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant
Number analyzed (Participants) | 9 | 15 | 13
Percentage of participants | 0 (0.0) [0.0 to 33.6] | 53.3 (26.6) [26.6 to 78.7] | 23.1 (5.0) [5.0 to 53.8]

54. Primary Outcome: Percentage of Participants Reporting SAEs From Vaccination 1 Through the Duration of the Study in Participants Aged >=5 to <12 Years
Description: as for outcome 53
Time Frame: From Vaccination 1 to 6 months after Vaccination 4 (approximately 14 months)
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant
Number analyzed (Participants) | 19 | 24 | 22
Percentage of participants | 15.8 (3.4) [3.4 to 39.6] | 20.8 (7.1) [7.1 to 42.2] | 13.6 (2.9) [2.9 to 34.9]

55. Primary Outcome: Percentage of Participants Reporting SAEs From Vaccination 1 Through the Duration of the Study in Participants Aged >=12 to <18 Years
Description: as for outcome 53
Time Frame: From Vaccination 1 to 6 months after Vaccination 4 (approximately 14 months)
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant
Number analyzed (Participants) | 7 | 1 | 7
Percentage of participants | 0 (0.0) [0.0 to 41.0] | 0 (0.0) [0.0 to 97.5] | 0 (0.0) [0.0 to 41.0]

56. Primary Outcome: Percentage of Participants Reporting SAEs From Dose 1 Through the Duration of the Study in Participants Aged >=18 Years
Description: as for outcome 53
Time Frame: From Vaccination 1 to 6 months after Vaccination 4 (approximately 14 months)
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
Number analyzed (Participants) | 5 | 1 | 1
Percentage of participants | 20.0 (0.5) [0.5 to 71.6] | 0 (0.0) [0.0 to 97.5] | 100.0 (2.5) [2.5 to 100.0]

ADVERSE EVENTS:
Time Frame: Local reactions/systemic events (systematic assessment): Day 1 to Day 7 after each dose. Non-systematic assessment: AEs were reported from Day 1 of dose 1 up to 1 month after dose 4 (approximately 9 months). For SAE, from Dose 1 on Day 1 to 6 months after Dose 4 (approximately 14 months).
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Some Adverse Events were collected in both systematic and non-systematic assessment methods.
Arm/Group | >=2 to <5 Years With Immunomodulatory Therapy | >=2 to <5 Years With Solid Organ Transplant | >=2 to <5 Years With Stem Cell Transplant | >=5 to <12 Years With Immunomodulatory Therapy | >=5 to <12 Years With Solid Organ Transplant | >=5 to <12 Years With Stem Cell Transplant | >=12 to <18 Years With Immunomodulatory Therapy | >=12 to <18 Years With Solid Organ Transplant | >=12 to <18 Years With Stem Cell Transplant | >=18 Years With Immunomodulatory Therapy | >=18 Years With Non-Small Cell Lung Cancer | >= 18 Years With Haemodialysis
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/15 | 0/13 | 0/19 | 0/24 | 0/22 | 0/7 | 0/1 | 0/7 | 0/5 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/9 | 8/15 | 3/13 | 3/19 | 5/24 | 3/22 | 0/7 | 0/1 | 0/7 | 1/5 | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 8/9 | 13/15 | 10/13 | 18/19 | 23/24 | 22/22 | 7/7 | 1/1 | 6/7 | 4/5 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | >=2 to <5 Years With Immunomodulatory Therapy (N=9) | >=2 to <5 Years With Solid Organ Transplant (N=15) | >=2 to <5 Years With Stem Cell Transplant (N=13) | >=5 to <12 Years With Immunomodulatory Therapy (N=19) | >=5 to <12 Years With Solid Organ Transplant (N=24) | >=5 to <12 Years With Stem Cell Transplant (N=22) | >=12 to <18 Years With Immunomodulatory Therapy (N=7) | >=12 to <18 Years With Solid Organ Transplant (N=1) | >=12 to <18 Years With Stem Cell Transplant (N=7) | >=18 Years With Immunomodulatory Therapy (N=5) | >=18 Years With Non-Small Cell Lung Cancer (N=1) | >= 18 Years With Haemodialysis (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | >=2 to <5 Years With Immunomodulatory Therapy (N=9) | >=2 to <5 Years With Solid Organ Transplant (N=15) | >=2 to <5 Years With Stem Cell Transplant (N=13) | >=5 to <12 Years With Immunomodulatory Therapy (N=19) | >=5 to <12 Years With Solid Organ Transplant (N=24) | >=5 to <12 Years With Stem Cell Transplant (N=22) | >=12 to <18 Years With Immunomodulatory Therapy (N=7) | >=12 to <18 Years With Solid Organ Transplant (N=1) | >=12 to <18 Years With Stem Cell Transplant (N=7) | >=18 Years With Immunomodulatory Therapy (N=5) | >=18 Years With Non-Small Cell Lung Cancer (N=1) | >= 18 Years With Haemodialysis (N=1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Donor specific antibody present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour necrosis factor receptor-associated periodic syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (HEADACHE) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 11 (25) | 11 (16) | 9 (17) | 7 (15) | 1 (1) | 6 (8) | 4 (9) | 1 (1) | 0 (0)
Amblyopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 2 (2) | 3 (4) | 2 (2) | 5 (8) | 5 (5) | 2 (4) | 2 (3) | 0 (0) | 2 (5) | 3 (6) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (VOMITING) (Gastrointestinal disorders) | 1 (1) | 3 (4) | 4 (4) | 2 (2) | 4 (5) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (NEW OR WORSENED JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (10) | 2 (2) | 3 (3) | 2 (4) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (NEW OR WORSENED MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 6 (10) | 8 (10) | 3 (3) | 3 (9) | 1 (1) | 3 (6) | 2 (5) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr viraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (CHILLS) (General disorders) | 2 (2) | 1 (1) | 1 (1) | 7 (9) | 3 (3) | 5 (7) | 5 (10) | 1 (1) | 1 (2) | 2 (5) | 0 (0) | 1 (1)
Erythema (REDNESS) (General disorders) | 3 (4) | 3 (5) | 0 (0) | 7 (10) | 5 (7) | 6 (13) | 3 (7) | 0 (0) | 2 (4) | 1 (2) | 0 (0) | 0 (0)
Fatigue (FATIGUE) (General disorders) | 3 (4) | 3 (3) | 3 (3) | 14 (34) | 17 (31) | 14 (31) | 6 (18) | 1 (2) | 5 (10) | 4 (11) | 1 (2) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 4 (6) | 3 (6) | 4 (4) | 16 (50) | 18 (43) | 19 (40) | 6 (20) | 1 (4) | 5 (12) | 4 (13) | 1 (3) | 1 (1)
Medical device site inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (FEVER) (General disorders) | 2 (3) | 1 (1) | 2 (2) | 2 (4) | 2 (2) | 5 (6) | 3 (7) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Swelling (SWELLING) (General disorders) | 1 (2) | 1 (2) | 1 (1) | 5 (8) | 4 (6) | 8 (17) | 2 (8) | 1 (1) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast enlargement (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT04895982/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT04895982/SAP_001.pdf